AnaptysBio Inc. Protocol No: ANB020-003 Version No.1.0 24 July 2019

# 16.1.9 Documentation of statistical methods

| Document | Date |
|----------------------------------------|------------------|
| Statistical Analysis Plan, Version 1.0 | 07 February 2018 |
| Table Shells, Version 1.0 | 07 February 2018 |
| Figure Shells, Version 1.0 | 07 February 2018 |
| Listing Shells, Version 1.0 | 07 February 2018 |



AnaptysBio Inc PROTOCOL ANB020-003 

# Statistical Analysis Plan

Study Number: ANB020-003

Placebo-Controlled Proof of Concept Study to Investigate ANB020 Activity in Adult Patients with Peanut Allergy

Author:

Version Number: Final 1.0

Date: 07 Feb 2018

\\lieedc-nas01a\\biosdata\\AnaptysBio\\ANB020\\CYA74393\\Biostatistics\\Documentation\\SAP\\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Protocol No: ANB020-003

24 July 2019

STATISTICAL ANALYSIS PLAN

AnaptysBio In PROTOCOL ANB020-00 Page 2 of

### Statistical Analysis Plan Signature Page

Statistical Analysis Plan Draft 2.0 (Dated 25Jul2017) for Protocol ANB020-003,

| | Name | Signature | Date |
|-----------|----------|-----------|---------|
| Author: | 3 | | мммүүүү |
| Position: | | | |
| Company: | IQVIA*** | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|------------------------------|---------|-----------|-----------|
| Reviewed and<br>Approved By: | | | DDMMNYYYY |
| Position: | - 7 | | |
| Company: | IQVIATM | | |
| Reviewed and<br>Approved By: | | | DDMMNYYYY |
| Position: | | | |
| Company: | IQVIATM | | |
| Reviewed and | | | DOMMMYYYY |
| | | | HAPR2018 |

Template No: C\$\_TP\_BS016 Revision 4 Effective Date: 01Apr2016

| STATISTICAL ANALYSIS | PLAN | Anapty<br>PROTOCOL ANBI<br>Pag |
|---|---|---|
| Position: | Medical Writer 1 | |
| Company: | IOVIATM | |
| Reviewed and<br>Approved By: | | DDMMMYYYY 12 A PP 201 |
| Position: | | |
| Company: | IQVIATM | A de la companya de l |
| Reviewed and<br>Approved By: | | DDMMMYYYY / / PATR ZOIS |
| Position: | | |
| Company: | AnaptysBio, Inc. | |
| ocument: Weeds-nas01a<br>ulhor: Preenan Sark | | Biostatistics\Documentation\\3AP\Final2018-0<br>Version Number. Final 1.0<br>Version Date: 07Feb2018 |


24 July 2019

€IQVIA

STATISTICAL ANALYSIS PLAN


# Statistical Analysis Plan Signature Page

Statistical Analysis Plan Draft 2.0 (Dated 25Jul2017) for Protocol ANB020-003.

| | Name | Signature | Date |
|-----------|---------|-----------|---------|
| Author: | | | MMMYYYY |
| Position: | | | |
| Company: | IQVIATM | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|--------------|---------|-----------|------------|
| Reviewed and | | | DDMMMYYYY |
| Approved By: | | | 11-4-18 |
| Position: | | | |
| Company: | IQVIATM | | |
| Reviewed and | | | DDMMMYYYY |
| Approved By: | | | |
| Position: | | | |
| Company: | IQVIATM | | |
| Reviewed and | | | DDMMMYYYY |
| Approved By: | | | 11APR 2018 |

Document: \text{Vicedo-nas01abiosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07\text{Version Number.}\text{Final 1.0\text{Version Date:}}\text{Version Date:}\text{Version Date:}

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016




# **List of Reviewers**

| Reviewer Name | Position/ Role | Company |
|---------------|----------------|------------------|
| | į | IQVIA™ |
| | | IQVIA™ |
| | | IQVIA™ |
| | | IQVIA™ |
| | | AnaptysBio, Inc. |

Document: Author: Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




# **Modification History**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from Previous Authorized Version |
|---|---|---|---|
| Draft 1.0 | 08 Mar 2017 | | Not Applicable – First ∀ersion |
| Version 1.0 | 16 Mar 2017 | | Addressed client comments |
| Draft 2.0 | 05 Jun 2017 | | Applied changes based on protocol amendment 2.0 dated 30May2017 |
| Draft 2.0 | 13 Jun 2017 | | Implemented SBR comments |
| Draft 2.0 | 28 Jun 2017 | | Implemented PK comments |
| Draft 2.0 | 25 Jul 2017 | | Implemented MW comments, changes based on protocol amendment 3.0 dated 30Jun2017 |
| Draft 3.0 | 07 Feb 2018 | | Implemented PK comments |
| Final Draft | 10 Apr 2018 | | Prepared the document for Sign off before DBL |

Document: Author: Version Number: Final 1.0 Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4



STATISTICAL ANALYSIS PLAN


# **Table of Contents**

| | RODUCTION | 11 |
|---|---|---|
| | IDY OBJECTIVES | |
| 2.1. | Primary Objectives | 11 |
| 2.2. | Secondary Objectives | 11 |
| 2.3. | Exploratory Objectives | 12 |
| | DY DESIGN | |
| 3.1. | General Description | |
| 3.2. | Schedule of Events | |
| | Scriedule of Events | 13 |
| 3.3. | Changes to Analysis from Protocol | |
| | NNED ANALYSIS | |
| 4.1. | Data Monitoring Committee (DMC) | |
| 4.2. | Interim Analysis | |
| 4.3. | Final Analysis | 14 |
| <ol><li>5. ANA</li></ol> | LYSIS SETS | 14 |
| 5.1. | All Patients Screened [SCR] | 14 |
| 5.2. | Randomized Analysis Set [RND] | |
| 5.3. | Full Analysis Set [FAS] | |
| 5.4. | Safety Analysis Set [SAF] | |
| 5.5. | Pharmacokinetic Analysis Set [PK] | |
| 5.6. | Pharmacodynamic Analysis Set [PD] | 15 |
| | IERAL CONS DERATIONS | 15 |
| 6.1. | Reference Start Date and Study Day | |
| 6.2. | Baseline | 17 |
| 6.3. | Retests, Unscheduled Visits and Early Termination Data | 17 |
| 6.4. | Windowing Conventions. | |
| 6.5. | Statistical Tests | 17 |
| 6.6. | Common Calculations | 18 |
| 6.7. | Software Version | 18 |
| | TISTICAL CONSIDERATIONS | 18 |
| 7.1. | Adjustments for Covariates and Factors to be Included in Analyses | 18 |
| 7.2. | Multicenter Studies | 10 |
| 7.3. | Missing data | |
| 7.4. | Multiple Comparisons/ Multiplicity | 10 |
| 7.5. | Number Companions Multiplicity | 10 |
| | Examination of Subgroups | |
| | PUT PRESENTATIONS | |
| | POSITION AND WITHDRAWALS | |
| | DEMOGRAPHIC AND OTHER BASEL NE CHARACTERISTICS | |
| 10.1. | Derivations | |
| 11. F | PROTOCOL DEVIATIONS | 20 |
| 12. | SURGICAL AND MEDICAL HISTORY | 21 |
| 13. ( | CONCOMITANT ILLNESSES | 21 |
| 14. ( | CONCOMITANT MEDICATIONS | 21 |
| | STUDY MEDICATION EXPOSURE | |
| | STUDY MEDICATION COMPLIANCE | |
| | FFICACY OUTCOMES | |
| 17.1. | Primary Efficacy | |
| 17.1.1. | PRIMARY EFFICACY ENDPOINT | |
| 17.1.1. | ANALYSIS OF PRIMARY EFFICACY ENDPOINT | 22 |
| 17.2. | Secondary Efficacy | |
| 17.2.1. | SECONDARY EFFICACY ENDPOINT | |
| 17.2.2. | SECONDARY PHARMACOKINETIC ENDPOINT | 23 |
| 17.2.3. | ANALYSIS OF SECONDARY EFFICACY ENDPOINT | 23 |
| 17.3. | Exploratory Efficacy | |
| 17.3.1. | EXPLORATORY EFFICACY ENDPO NTS | |
| 17.3.2. | EXPLORATORY PHARMACODYNAMICS ENDPO NTS | 24 |
| 17.3.3. | ANALYSIS OF EXPLORATORY EFFICACY ENDPO NTS | |
| 18. 5 | | 25 |

Version Number: Final 1.0 Author: Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Document:

Version No.1.0

Protocol No: ANB020-003 24 July 2019



## AnaptysBio Inc PROTOCOL ANB020-003 

# STATISTICAL ANALYSIS PLAN

| 18.1. | Adverse Events | 25 |
|---------------|---------------------------------------|----|
| 18.2. | Deaths | 26 |
| 18.3. | Laboratory Evaluations | 26 |
| 18.4. | ECG Evaluations | 27 |
| 18.4.1. | ECG SPECIFIC DERIVATION | 27 |
| 18.4.2. | ECG MARKEDLY ABNORMAL CRITERIA | 28 |
| 18.5. | Vital Signs | 28 |
| 18.6. | Physical Examination | 28 |
| 18.7. | Other Safety Assessments (Spirometry) | 28 |
| | PHARMACOK NETIC OUTCOMES | 29 |
| 20. F | PHARMACODYNAMIC OUTCOMES | 31 |
| 21. ( | GENETIC ANALYSIS | 32 |
| <b>22</b> . [ | OATA NOT SUMMARIZED OR PRESENTED | 32 |
| 23. F | REFERENCES | 33 |
| <b>APPEND</b> | IX 1. Partial Date Conventions | 33 |
| TURE 1: Sc | hematic of Study Design | 13 |

Document: \\ieedc-nas01a\\biosdata\\AnaptysBio\\ANB020\\CYA74393\\Biostatistics\\Documentation\\SAP\\Final2018-02-\overline{07} \
Author: \quad \text{Version Number: Final 1.0} \quad \text{Version Date: 07Feb2018}

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016




# List of Abbreviations and Definitions of Terms

| Abbreviation | Definition |
|---|---|
| AE | Adverse event |
| ANCOVA | Analysis of covariance |
| %AUC <sub>ex</sub> | Percentage of AUC <sub>(0-inf)</sub> obtained by extrapolation |
| AUC <sub>(0-inf)</sub> | Area under the concentration-time curve from time zero (predose) extrapolated to infinite time |
| AUC <sub>(0-last)</sub> | Area under the concentration-time curve from time zero (predose) to time of last quantifiable concentration |
| BLQ | Below the lower limit of quantitation |
| ВМІ | Body mass index |
| BP | Blood pressure |
| BPCFC | Blind placebo-controlled food challenge |
| CI | Confidence interval |
| CL | Systemic clearance following intravenous dosing |
| C <sub>max</sub> | Maximum observed concentration |
| CV | Coefficient of variation |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |

Document: Author: Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005



# STATISTICAL ANALYSIS PLAN


| EOS | End of Study |
|-----------------|----------------------------------------------|
| ET | Early Termination |
| gCV | Geometric coefficient of variation |
| Gmean | Geometric mean |
| HR | Heart rate |
| ICH | International Council for Harmonisation |
| IP | Investigational product |
| IV | Intravenous(ly) |
| λz | Apparent terminal rate constant |
| LLOQ | Lower limit of quantitation |
| LS | Least-squares |
| MedDRA | Medical Dictionary for Regulatory Activities |
| n | Sample size or number of observations |
| OFC | Oral Food Challenge |
| PD | Pharmacodynamic(s) |
| PK | Pharmacokinetic(s) |
| R <sub>sq</sub> | Coefficient of determination |
| SAE | Serious adverse event |

Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005



# STATISTICAL ANALYSIS PLAN


| SAP | Statistical analysis plan |
|---|---|
| SAS | Statistical analysis system |
| SD | Standard deviation |
| SI | System International |
| TEAE | Treatment emergent adverse event |
| t <sub>1/2</sub> | Apparent terminal half-life |
| tmax | Time to maximum observed concentration |
| Vss | Volume of distribution at steady state following intravenous dosing |
| Vz | Volume of distribution |
| WBC | White blood cell |
| WHO DD | World Health Organization Drug Dictionary |

Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4




#### 1. Introduction

This document describes the statistical analyses to be performed and data presentations to be produced for this phase II, randomized, double-blind, placebo-controlled, study to evaluate the safety, tolerability and efficacy of single IV infusion of 300 mg ANB020 in 20 Adult Patients with Peanut Allergy.

The purpose of this statistical analysis plan (SAP) is to ensure the credibility of the study findings by specifying the statistical approaches to the analysis of the double-blind data prior to database lock. This SAP was developed based on the International Conference on Harmonization (ICH) E3 and E9 Guidelines and in reference to the following document:

Protocol AnaptysBio ANB020-003 amendment 3 dated 30Jun2017.

Any deviations during the analysis and reporting process from the current SAP will be described and justified in the final report. Analysis issues that suggest changes to the principal features stated in the protocol will be documented in a protocol amendment. Otherwise, the SAP will be updated through an amendment with the changes in the analysis documented in the amendment.

#### 2. STUDY OBJECTIVES

#### 2.1. PRIMARY OBJECTIVES

To assess the safety and tolerability of single dose administration of ANB020 in adult patients with peanut allergy

To measure the response of adult patients with peanut allergy on Day 14 following an oral blind placebocontrolled food challenge (BPCFC) threshold and total cumulative peanut dose tolerated after administration of ANB020 or placebo compared to cumulative baseline peanut BPCFC

#### 2.2. SECONDARY OBJECTIVES

To compare the symptoms to peanut antigen challenge on Day 14 using the Oral Food Challenge (OFC) Symptoms Scoring Assessment Tool after administration of ANB020 or placebo compared to baseline peanut BPCFC symptoms

To describe the limited pharmacokinetics (PK) of ANB020 following a single, intravenous (IV) dose

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4




#### 2.3. EXPLORATORY OBJECTIVES

To assess the effect of ANB020 on circulating serum cytokines

To assess the effect of ANB020 on leukocytes within whole blood

To compare the immune response of ANB020 to placebo dosed patients in the ex vivo peanut antigen challenge

To measure the response of adult patients with peanut allergy on Day 45 following an oral BPCFC threshold and cumulative peanut dose tolerated after administration of ANB020 or placebo compared to cumulative baseline peanut BPCFC

To compare the symptoms to peanut antigen challenge on Day 45 using the OFC Symptoms Scoring Assessment Tool after administration of ANB020 or placebo compared to baseline peanut BPCFC symptoms

#### 3. STUDY DESIGN

#### 3.1. GENERAL DESCRIPTION

This is a Phase II, double-blind, placebo-controlled, proof of concept study to assess the safety and tolerability of ANB020 in adult patients with peanut allergy. This study will also investigate the effects of ANB020 or placebo in adult peanut allergic patients following an oral BPCFC at 2 and 6 weeks post ANB020 or placebo administration. The effects of ANB020 on the immune response to peanut upon ex vivo peanut antigen challenge will be evaluated.

No formal statistical calculation has been performed for sample size. Approximately 20 patients will be enrolled in the study.

Patients will be randomized in a 3:1 ratio to receive ANB020 (300 mg/100 mL) or matching 100 mL placebo (0.9% sodium chloride) administered through intravenous route.

A schematic of the study design is included as Figure 1:

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document:

Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




Figure 1: Schematic of Study Design



#### 3.2. SCHEDULE OF EVENTS

The schedule of events can be found in Section 4.1, Table 4.1 of the protocol

Document: \\ieedc-nas01a\\biosdata\\AnaptysBio\\ANB020\\CYA74393\\Biostatistics\\Documentation\\SAP\\Final2018-02-\\0007\\Author: \quad \qquad \quad \qquad \quad \quad

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

15




#### 3.3. CHANGES TO ANALYSIS FROM PROTOCOL

No changes from the analysis planned in the protocol were made.

### 4. PLANNED ANALYSIS

This SAP describes the methodology for final analysis.

### 4.1. DATA MONITORING COMMITTEE (DMC)

No DMC is planned of this study.

#### 4.2. INTERIM ANALYSIS

No interim analysis is planned for this study.

#### 4.3. FINAL ANALYSIS

All final, planned statistical analyses identified in this SAP will be performed by the IQVIA Biostatistics department.

Analysis of the PK and pharmacodynamics (PD) of ANB020 and the associated figures, will be the responsibility of the clinical pharmacokineticist (PK analyst) at IQVIA. The PK/PD summaries and data listings will be the responsibility of the ECD biostatistician at IQVIA.

### 5. ANALYSIS SETS

Summaries will be presented by treatment and overall as appropriate.

Listings will be presented for all patients available in the data transfer received from data management.

The following analysis sets will be used:

# 5.1. ALL PATIENTS SCREENED [SCR]

Patients who have signed the informed consent form and have been screened.

#### 5.2. RANDOMIZED ANALYSIS SET [RND]

All patients who have been allocated to a randomized treatment arm, regardless of whether they received the planned treatment or not. Patients will be considered according to their randomized

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




treatment.

## 5.3. FULL ANALYSIS SET [FAS]

All patients who have received ANB020 or placebo and were present in the study until Day 14 with post baseline BPCFC and OFC results present. The full analysis set will be used for all efficacy analyses. Patients will be considered according to their randomized treatment.

#### 5.4. SAFETY ANALYSIS SET [SAF]

All patients who have received any portion of ANB020 or placebo infusion. The safety analysis set will be used for all safety analyses. Patients will be considered according to their actual treatment received.

# 5.5. PHARMACOKINETIC ANALYSIS SET [PK]

All patients who have received ANB020 and have at least one post dose serum concentration data value available for ANB020 without any events or protocol deviation deemed to affect PK assessments. The PK analysis set will be used for all PK analyses.

#### 5.6. PHARMACODYNAMIC ANALYSIS SET [PD]

All patients who have received at least one dose of ANB020 or placebo and provide at least one evaluable post dose PD measurement without any events or protocol deviation deemed to affect PD assessment. The PD analysis set will be used for all PD analyses.

#### 6. GENERAL CONSIDERATIONS

The following descriptive statistics will be presented in summary tables:

Continuous variables: will be summarized by treatment group using number of valid cases (n), mean, median, standard deviation (SD), minimum, and maximum.

Categorical variables: will be summarized by treatment group using frequency tables [frequencies (n) and percentages (%)]. Percentages are routinely based on the total category count excluding the missing category if not otherwise mentioned. Missing category with zero count will not be presented.

In general, for non-PK/PD data, the number of decimal places displayed for each statistic will be determined as follows:

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Author:




Mean and median: 1 more than the number of decimal places allotted in the raw data received from data management.

Standard deviation: 2 more than the number of decimal places allotted in the raw data.

Minimum and maximum: equal to the number of decimal places allotted in the raw data.

Percentages: All percentages between 0 and 100 will be rounded to one decimal unless there is a need to report more than one decimal for percentages.

Ranges will be reported to the same number of decimal places displayed by the laboratory.

P-values, if any, shall be reported to four decimal places or as <0.0001.

Pharmacokinetic parameters will be rounded for reporting purposes both in the summary tables and by-subject listings. For the calculation of descriptive statistics and the statistical analysis, rounded values as presented in the data listings will be used. All data will be reported and analyzed with the same precision as the source data regardless of how many significant figures or decimals the data carry. For most derived PK parameters, 3 significant digits will be used as the standard rounding procedure, with the following exceptions:

Parameters directly derived from source data [e.g., maximum observed concentration (C<sub>max</sub>)] will be reported and analyzed with the same precision as the source data.

Parameters derived from actual elapsed sample collection times [e.g., time to maximum observed concentration (t<sub>max</sub>)] will be reported in hours with 2 decimal places.

Apparent terminal rate constant ( $\lambda_z$ ) will be reported with 4 decimal places.

For PK data, reporting of mean (arithmetic and geometric), SD, and median will carry 1 more significant figure than the source data. Minimum and maximum will carry the same number of significant figures as the source data. The bounds of any confidence intervals (CIs) will be reported with 2 decimals, and coefficient of variation (CV) will be reported as a percentage to 1 decimal place.

Extra measurements (such as unscheduled or repeat assessments) will not be included in the descriptive statistics, but will be included in subject listings. Pharmacokinetic summaries will be presented for all subjects in the PK analysis set as defined in Section 5.5. Similarly, PD summaries will be presented for all subjects in the PD analysis set as defined in Section 5.6. Data from subjects excluded from an analysis set will be included in the data listings, but not in the summaries.

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Author:



STATISTICAL ANALYSIS PLAN


### 6.1. REFERENCE START DATE AND STUDY DAY

The reference start date is defined as the day of the first dose of study medication (Day 1 is the day of the first dose of study medication), and will appear in every listing where an assessment date or event date appears.

The study day will be calculated from the reference start date, and will be used to show start/stop day of assessments and events.

If the date of the event is on or after the reference date then:

Study Day = (date of event - reference date) + 1

If the date of the event is prior to the reference date then:

Study Day = (date of event – reference date)

If the event date is partial or missing, Study Day, and any corresponding durations will appear partial or missing in the listings.

Refer to Appendix 1 for more details.

### 6.2. BASELINE

The nearest non-missing measurements taken prior to ANB020 or placebo administration, i.e., reference start date, will be considered as baseline. If the last non-missing measurement and the reference start date coincide, that measurement will be considered baseline, but Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline.

### 6.3. RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

Listings will include scheduled, unscheduled, retest, and early discontinuation data.

#### 6.4. WINDOWING CONVENTIONS

Not applicable.

### 6.5. STATISTICAL TESTS

All tests of treatment effects will be conducted at a 2-sided alpha level of 0.05, or with 2-sided 95% CIs.

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Author: Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005



STATISTICAL ANALYSIS PLAN


#### 6.6. COMMON CALCULATIONS

For quantitative measurements, change from baseline will be calculated as:

Test Value at Visit X - Baseline Value

#### 6.7. SOFTWARE VERSION

All analyses will be conducted using SAS System® Version 9.2 or higher.

The non-compartmental PK analysis will be conducted using SAS System® and/or Phoenix WinNonlin® 6.4 or higher, and PK graphics will be prepared using SigmaPlot® 12.5, or higher.

#### 7. STATISTICAL CONSIDERATIONS

#### 7.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The change from baseline on Day 14 of tolerated peanut dose will be compared between ANB020 and placebo using an analysis of covariance (ANCOVA) with treatment as fixed effect and baseline results as a covariate. Similarly, the mixed model for repeated measures for analysis of exploratory endpoints will include baseline and baseline by visit terms as covariates.

# 7.2. MULTICENTER STUDIES

Not applicable as this is a single center study.

#### 7.3. MISSING DATA

No imputations will be performed on missing data.

### 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

Not applicable.

### 7.5. EXAMINATION OF SUBGROUPS

No subgroups analysis will be performed for this study.

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4




# 8. OUTPUT PRESENTATIONS

The templates provided with this SAP describe the presentations for this study and the format and content of the summary tables, figures, and listings are to be provided by IQVIA Biostatistics.

All visit assessments will be presented according to the nominal visit name.

#### 9. DISPOSITION AND WITHDRAWALS

All patients who provide informed consent will be accounted.

Data collected in Early Termination (ET) and End of Study (EOS) pages in the electronic Case Report Form (eCRF) will be used to present disposition and withdrawal results. Frequency table will be provided for:

number of patients in the All Patients Screened Set (provided informed consent and demographic details available)

number of patients eligible at screening

number of patients eligible at Day 1

number of screen failures

number of patients in the Randomized Analysis Set

number of patients administered the treatment

number of patients in the Full Analysis Set

number of patients in the Safety Analysis Set

number of patients in the Pharmacokinetic Analysis Set

number of patients in the Pharmacodynamic Analysis Set

number of patients who discontinued the study

primary reason for discontinuation

number of patients who completed the study

A listing will be presented with the following details.

screening date

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4



STATISTICAL ANALYSIS PLAN


assigned treatment

screen failure (Yes/No)?

completed study (Yes/No)?

If not completed the study, then reason for discontinuation

A separate listing will be presented of eligibility criteria deviations for which the all patient screened population will used.

# 10. Demographic and other Baseline Characteristics

Demographic data and other baseline characteristics will be presented for the Randomized Analysis Set. No statistical testing will be carried out for demographic or other baseline characteristics.

Summary statistics will be provided for:

Age (years) - calculated relative to date of consent

Weight (kg)

Height (cm)

BMI (kg/m<sup>2</sup>)

Frequency tables will be provided for:

Gender

Ethnicity

Race

A listing for patient demographic data and other baseline characteristics will be presented.

#### 10.1. **DERIVATIONS**

BMI  $(kg/m^2)$  = weight (kg)/ height  $(m)^2$ 

## 11. PROTOCOL DEVIATIONS

All protocol deviations observed during study conduct will be captured in Clinical Trial Management System (CTMS).

Document: Author:

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




The Investigator and Sponsor will review the protocol violation records from CTMS and provide confirmation on the categorization of violations as major or other.

Major protocol deviations or events include changes to the procedures that may impact the quality of the data or any circumstances that can alter the evaluation of the PK data. Examples include, but may not be limited to, sample processing errors that lead to inaccurate bioanalytical results, incomplete dose administered, incomplete PK profile collected, use of disallowed concomitant medication thought to affect PK. In the case of a major protocol deviation or event, affected PK data collected will be excluded from the summaries and statistical analyses, but will still be reported in the study result listings.

A frequency table for major protocol violations will be provided for Randomized Analysis Set. Major protocol deviations or events that impact the quality of the PK and/or PD data will be listed only.

A list of major protocol deviations that involve eligibility criteria or could significantly affect study assessments will be provided. The incidence of each protocol violation will be listed.

#### 12. SURGICAL AND MEDICAL HISTORY

Frequency tables will be provided for medical history findings summarized by body system for the Randomized Analysis Set. Version 19.1 of Medical Dictionary for Regulatory Activities (MedDRA) will be used.

AEs due to BPCFC at screening visit will be captured as medical history.

A listing of medical history diagnoses with all details will be presented.

### 13. CONCOMITANT ILLNESSES

Not applicable.

### 14. CONCOMITANT MEDICATIONS

A frequency table will be provided for concomitant medications and will be summarized by Anatomic, therapeutic and chemical classification (ATC) Level 1 and 3 for Safety Analysis Set. Concomitant medication will be coded using WHO drug dictionary Version Dec 2016.

See Appendix 1 for handling of partial dates for medications. If it is not possible to define a medication as prior, concomitant, or post treatment, the medication will be classified by the worst case; i.e.,

\\lieedc-nas01a\\biosdata\\AnaptysBio\\ANB020\\CYA74393\\Biostatistics\\Documentation\\SAP\\Final2018-02-07 Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016

Document:

Author:



STATISTICAL ANALYSIS PLAN


concomitant.

'Prior' medications are medications which started and stopped prior to the first dose of study medication.

'Concomitant' medications are medications which:

- started prior to, on or after the first dose of study medication,
- AND ended on or after the date of first dose of study medication or were ongoing at the end of the

A listing for medication with all details will be presented and safety analysis set will be used for the

# 15. STUDY MEDICATION EXPOSURE

A listing of exposure to Investigational Product will be presented, with details of start and end time of infusion, interruptions, and total volume administered. IP Administration data will be used to generate the listing.

# 16. STUDY MEDICATION COMPLIANCE

Overall compliance is expected as the study medication is being administered at the clinic, however no summary will be provided for compliance.

### 17. EFFICACY OUTCOMES

#### 17.1. **PRIMARY EFFICACY**

### 17.1.1. PRIMARY EFFICACY ENDPOINT

The difference in total cumulative tolerated peanut dose during BPCFC between post-treatment and baseline, following treatment with ANB020 or placebo on Day 14.

#### 17.1.2. ANALYSIS OF PRIMARY EFFICACY ENDPOINT

The null hypothesis for the primary efficacy analysis is:

H0: There is no difference in change from baseline on day 14 for total cumulative tolerated peanut dose during BPCFC between ANB020 and placebo.

Document: Author:

\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Version Number: Final 1.0

Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016



STATISTICAL ANALYSIS PLAN


Vs the alternative:

H1: There is a difference in change from baseline on day 14 for total cumulative tolerated peanut dose during BPCFC between ANB020 and placebo

The primary efficacy analysis will be carried out for the FAS population.

The actual and change from baseline values of primary efficacy endpoints will be summarized using appropriate descriptive statistics by treatment at all time points where assessment is done. Change from baseline will be evaluated where possible.

Regarding the primary efficacy endpoint, change from baseline on day 14 of tolerated dose will be compared between ANB020 and placebo using an ANCOVA with treatment as fixed effect and baseline results as a covariate.

The following statistics will be presented:

- Treatment difference 0
- Standard error of treatment difference 0
- 95% CI 0
- p-value o

The treatment difference and 95% CI will also be presented graphically.

Patient-wise data listings will be provided.

#### 17.2. SECONDARY EFFICACY

#### 17.2.1. SECONDARY EFFICACY ENDPOINT

Clinical scores of OFC Symptom Scoring Assessment Tool on Day 14

#### 17.2.2. SECONDARY PHARMACOKINETIC ENDPOINT

Maximum observed concentration (Cmax)

Time to maximum observed concentration (t<sub>max</sub>)

# 17.2.3. ANALYSIS OF SECONDARY EFFICACY ENDPOINT

The analysis of the secondary efficacy endpoint will be carried out in the similar way as of primary efficacy endpoint for FAS population.

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Author: Version Number: Final 1.0 Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4




For analysis of secondary PK endpoints, refer to Section 19 for details.

#### 17.3. **EXPLORATORY EFFICACY**

#### 17.3.1. EXPLORATORY EFFICACY ENDPOINTS

The difference in total cumulative tolerated peanut dose during BPCFC between post-treatment and baseline, following treatment with ANB020 or placebo on Day 45

Clinical scores of OFC Symptom Scoring Assessment Tool on Day 45

#### 17.3.2. EXPLORATORY PHARMACODYNAMICS ENDPOINTS

Serum cytokines will be evaluated including, but not be limited to, IL-4, IL-5, IL-9, IL-13, IL-33, and sST2

Differential white blood cell counts (WBC) in the whole blood will be measured to monitor circulating leukocyte populations

For the ex vivo peanut antigen challenge, the whole blood peanut response assay will measure the cytokine levels released from pathogenic T cells

#### 17.3.3. ANALYSIS OF EXPLORATORY EFFICACY ENDPOINTS

The Full Analysis Set will be used for the efficacy analysis.

The actual and change from baseline values of all the exploratory endpoints will be summarized using appropriate descriptive statistics by treatment at all time points where assessment is done. Change from baseline will be evaluated where possible.

Change from baseline on day 45 for tolerated dose and OFC symptom scores will be compared between ANB020 and placebo using a mixed model for repeated measures with treatment, visit, and treatment by visit interaction as fixed effect, and baseline and baseline by visit terms as covariates. The data collected at baseline, day 14, and day 45 will be used in the model.

The following statistics will be presented:

- Treatment differences 0
- Standard error of treatment difference 0
- 95% CI 0
- p-value 0

Document: Author:

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07

Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




An appropriate covariance matrix (e.g., unstructured [UN]) will be used in the model.

The treatment difference and 95% CI will also be presented graphically.

Patient-wise data listings will be provided.

For analysis of exploratory PD endpoints, refer Section 20 for details.

#### 18. SAFETY OUTCOMES

Safety outcomes will be based on the Safety Analysis Set defined in Section 6.

There will be no statistical comparisons between the treatment groups for safety data.

#### 18.1. ADVERSE EVENTS

Adverse Events (AEs) will be coded using MedDRA Version 19.1.

Treatment emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or after the date and time of the IP infusion or if the event represents an exacerbation of a condition observed pre-treatment. This excludes AEs due to BPCFC. AEs due to BPCFC during screening visit will be captured in medical history events.

Non treatment emergent adverse event (Non-TEAE) will be defined as any AE that started after the informed consent form has been signed and before the first dose of study medication and did not qualify for TEAE in terms of severity.

Adverse events with missing start dates will be considered treatment-emergent. AEs with missing stop dates or with stop dates after the end of the study date will be considered to have been ongoing at the end of the study.

The relationship to investigational product will be presented as "Related" versus "Not Related". Here the relationship categories "Unrelated" and "Unlikely" collected in the eCRF will be mapped to "Not Related", while the categories "Possible", "Probable" and "Unknown" will be mapped to "Related".

For each treatment, numbers of events, patients experiencing adverse events and percentage will be tabulated. The following summary tables will be provided by system organ class and preferred term for each treatment group:

number of patients with at least one TEAE

number of patients with at least one serious TEAE

Document: Author:

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




# STATISTICAL ANALYSIS PLAN

- number of patients with at least one TEAE by severity 0
- number of patients with at least one TEAE by relationship to IP 0
- number of patients with at least one TEAE leading to discontinuation from the study 0
- number of patients with at least one TEAE leading to interruption of IP
- number of patients with at least one TEAE leading to death 0
- number of patients with non-TEAE
- number of patients with AEs due BPCFC

When calculating the number of patients who experience an AE, an event that occurred one or more times on treatment will contribute one observation to the numerator and denominator for all safety patients exposed to ANB020 or placebo for the respective treatment, i.e., the event will be counted only once per SOC and per PT with highest severity and worst relationship with IP.

Listings will be provided for TEAEs, Serious TEAEs, TEAEs leading to discontinuation from study or of IP, and TEAEs leading to deaths for safety analysis set.

#### 18.2. **DEATHS**

The number of patients with at least one TEAE leading to death will be summarized and listed as described above.

#### 18.3. LABORATORY EVALUATIONS

Results from both the central and local laboratory will be included in the reporting. Central laboratory results will be reported for hematology, clinical chemistry and urinalysis. Local urine pregnancy test results will be reported as well. The actual and change from baseline values for each laboratory parameter will be summarized using descriptive statistics (n, mean, SD, median, and range) by treatment and all available visits.

The following summaries will be provided for laboratory data:

- Incidence of abnormal values according to normal range criteria 0
- Potential clinical significance of clinical laboratory assessments

A shift table will be presented of the potential shifts from baseline to the final measurement of values that are clinically relevantly high or low.

A listing of patients with abnormal values or clinically significant changes will be presented.

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4



STATISTICAL ANALYSIS PLAN


Hematology and clinical laboratory data will be reported in System International (SI) units.

#### 18.4. **ECG EVALUATIONS**

The following ECG parameters will be summarized:

- Heart Rate (bpm)
- PR Interval (msec) 0
- QRS Interval (msec) 0
- QT Interval (msec) 0
- QTcB (msec) {based on Bazett formula} 0
- QTcF (msec) {based on Fridericia formula} 0

The actual and change from baseline values for the above parameters will be summarized using descriptive statistics (n, mean, SD, median, and range) by treatment and all available visits.

The overall assessment of ECG will be summarized using frequency and percentage of the following indications:

- Normal
- 0 Abnormal, Not Clinically Significant (ANCS)
- Abnormal, Clinically Significant (ACS) 0

A listing of ECG parameters and of the overall assessment will be provided.

### 18.4.1. ECG SPECIFIC DERIVATION

Bazett's Correction (msec)

$$QTcB \text{ (msec)} = \frac{QT \text{ (ms)}}{\sqrt{RR \text{ (ms)}/1000}}$$

Fridericia's Correction (msec)

$$QTcF \text{ (msec)} = \frac{QT \text{ (ms)}}{\sqrt[2]{RR \text{ (ms)}/1000}}$$

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Author:

Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005



STATISTICAL ANALYSIS PLAN


#### 18.4.2. ECG MARKEDLY ABNORMAL CRITERIA

Absolute values of the QT interval will be classified as:

- o >=450 msec
- o >=480 msec
- o >=500 msec

The change from Baseline of QT interval will be classified as:

- o >30 msec increase from baseline
- >60 msec increase from baseline

#### 18.5. VITAL SIGNS

The following Vital Signs measurements will be reported for this study:

- Blood Pressure (mmHg)
- Respiratory Rate (resp/min) 0
- Pulse Rate (breaths/min) 0
- Temperature (°C or °F)

The actual and change from baseline values for the above parameters will be summarized using descriptive statistics (n, mean, SD, median, and range) by treatment and all available visits.

A listing of the above parameters will be provided.

#### 18.6. PHYSICAL EXAMINATION

The frequency and percentage of patients with physical examination assessments will be summarized by body system and treatment group at each available visit.

A listings of physical examination findings will be provided.

#### 18.7. OTHER SAFETY ASSESSMENTS (SPIROMETRY)

For patients with a history of asthma, the following spirometry or peak flow parameters will be summarized for observed and change from baseline values by treatment group at each available visit:

Actual FEV1

Predicted FEV1

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




#### Percent Predicted

A detailed listing will be presented for spirometry.

# 19. PHARMACOKINETIC OUTCOMES

Pharmacokinetic analysis of the plasma concentration data for ANB020 will be performed at IQVIA, Overland Park, Kansas, United States. The actual sampling times will be used in the PK parameter calculations, and PK parameters will be derived using standard non-compartmental methods using Phoenix WinNonlin® 6.4 or higher (Pharsight Corp., Certara Company, Princeton, New Jersey, United States); and/or SAS® Version 9.2 or higher. Graphics may be prepared with SAS® Version 9.2, or higher; SigmaPlot® 12.5, or higher (Systat Software, Inc., San Jose, California, United States); or Phoenix WinNonlin® 6.4, or higher.

A listing of PK blood sample collection times as well as derived sampling time deviations will be provided. A subject listing of all concentration-time data for ANB020 will be provided.

Concentration data of ANB020 will be summarized by treatment and nominal time point using the number of observations (n), and number of observations ≥ lower limit of quantitation (LLOQ), arithmetic mean, SD, CV, minimum, median, and maximum. Concentrations below the lower limit of quantitation (BLQ) will be treated as zero for calculation of descriptive statistics. If the calculated mean concentration is BLQ, the mean value will be reported as BLQ and the SD and CV will be reported as not applicable (NA). Missing data will not be interpolated. If 1 or more concentrations at a given time point are missing, they will be reported as missing and will be omitted from the calculation of descriptive statistics.

Plots of the mean plasma concentration-time profile for ANB020 will be presented by nominal sampling time on linear and semi-logarithmic scales. Individual concentration-time data will be listed and plotted by actual sampling times on linear and semi-logarithmic scales.

For the calculation of PK parameters, concentrations that are BLQ will be assigned a value of zero if they precede quantifiable samples prior to t<sub>max</sub>. Any anomalous concentration values observed at predose will be identified in the study report and will be used for the computation of PK parameters if the anomalous value is not greater than 5% of C<sub>max</sub>. If the anomalous value is greater than 5% of C<sub>max</sub>, the PK parameters for the given subject will be included in listings but excluded from summary presentations and analyses. Following Cmax, BLQ values embedded between 2 quantifiable data points will be treated

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005




### STATISTICAL ANALYSIS PLAN

as missing. Trailing BLQ values (BLQ values after the last quantifiable concentration) will be set to zero. If consecutive BLQ concentrations are followed by quantifiable concentrations in the terminal portion of the concentration curve, these quantified values will be excluded from the PK analysis by setting them to missing.

The following PK parameters will be computed for ANB020, if data permits:

| C <sub>max</sub> | Maximum concentration in serum (µg/mL), obtained directly from the observed concentration versus time data. |
|---|---|
| t <sub>max</sub> | Time of maximum concentration (h), obtained directly from the observed concentration versus time data. |
| AUC <sub>(0-inf)</sub> | Area under the concentration-time curve in serum from time zero (predose) extrapolated to infinite time (h· $\mu$ g/mL), calculated by linear up/log down trapezoidal summation and extrapolated to infinity by addition of the last quantifiable concentration divided by the apparent terminal rate constant: $AUC_{(0-last)} + C_{last}/\lambda_z.$ |
| AUC <sub>(0-last)</sub> | Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration ( $h\cdot \mu g/mL$ ), calculated by linear up/log down trapezoidal summation. |
| CL | Systemic clearance (L/h), calculated as dose/ AUC <sub>(0-inf)</sub> . |
| λz | Apparent terminal rate constant (1/h), determined by linear regression of the terminal points of the log-linear concentration-time curve. |
| t <sub>1/2</sub> | Apparent terminal half-life (h), determined as (ln2/ $\lambda z$ ). |
| V <sub>ss</sub> | Volume of distribution at steady state following intravenous dosing (L), calculated as mean residence time (extrapolated to infinity) multiplied by systemic clearance. |
| Vz | Volume of distribution (L), estimated by dividing the systemic clearance by |

Document: Author:

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07

Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016




λz.

The following ANB020 PK parameters will be calculated for diagnostic purposes and listed, but will not summarized:

| λz_lower | Start time (h) of the log-linear regression to determine $\lambda_Z$ and $t_{1/2}$ . |
|---|---|
| λz_upper | End time (h) of the log-linear regression to determine $\lambda_Z$ and $t_{1/2}.$ |
| t <sub>1/2</sub> , Interval | The time interval (h) of the log-linear regression to determine $\lambda_Z$ and $t_{1/2}$ , calculated as $\lambda_Z$ _upper – $\lambda_Z$ _lower, |
| t <sub>1/2</sub> , N | Number of data points included in the log-linear regression analysis used to calculate $\lambda_Z$ and $t_{1/2}$ . A minimum of 3 data points is required. |
| R <sub>sq</sub> | Coefficient of determination for calculation of $\lambda_Z$ . A minimum of 3 data points (excluding $C_{max}$ ) will be used for determination of the terminal linear phase of the concentration-time profile. If the Rsq is less than 0.800 then $\lambda_Z$ , $t_{1/2}$ , $AUC_{(0-inf)}$ , $CL$ , $V_{ss}$ , and $V_Z$ will be listed but not included in summary presentations or analyses. |
| %AUC <sub>ex</sub> | Percentage of AUC <sub>(0-inf)</sub> obtained by extrapolation, calculated as [( $C_{last}/\lambda z$ )/ AUC <sub>(0-inf)</sub> ×100]. If the extrapolated area is greater than 20.0% of AUC <sub>(0-inf)</sub> , then AUC <sub>(0-inf)</sub> will listed but not included in summary presentations or analyses. |

The PK parameters, with the exception of t<sub>max</sub>, will be summarized by treatment using n, arithmetic mean, SD, CV, minimum, median, maximum, geometric mean (Gmean), and geometric CV (gCV). The PK parameter t<sub>max</sub> will be reported with n, minimum, median, and maximum only.

# 20. PHARMACODYNAMIC OUTCOMES

The PD analysis set will be used for PD analysis.

Observed values, change from baseline and relative change from baseline for circulating cytokines,

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4

Effective Date: 01Apr2016




differential WBC counts (circulating leukocytes), and cytokine levels released from pathogenic T-cells (ex vivo whole blood peanut response assay) will be summarized with descriptive statistics including 95% CIs for the mean by nominal time point and treatment. Relative change from baseline is calculated as (actual-baseline)/baseline and will be reported as percentage.

Comparison between ANB020 and placebo will be performed using a repeated measures ANCOVA model on observed values with treatment, time point of measurement, and treatment by time point interaction as fixed effects, and baseline value as a covariate. An unstructured covariance matrix will be used. If the model fails to converge, then appropriate covariance matrix (e.g., compound symmetric) will be selected based on Akaike Information Criteria (AIC). All tests of treatment effects will be conducted at a 2-sided alpha level of 0.05 or with 2-sided 95% CIs. The following statistics will be presented:

- Least-squares (LS) mean for treatment difference 0
- Standard error of LS mean of difference 0
- 95% CI for LS mean treatment difference 0
- p-value for comparison of ANB020 versus placebo

Log or other transformation may be applied upon specific parameters as appropriate to meet the analysis assumptions.

A listing of PD blood sample collection date and times will be provided. A subject listing of all PD data (serum cytokines IL-4, IL-5, IL-9, IL-13, IL-33 and sST2, leukocytes in whole blood, and cytokine levels released from pathogenic T-cells following the ex vivo whole blood peanut response assay) will be provided. All PD parameters will be summarized as described in Section 6, General Considerations, and observed values will be presented graphically in scatter plots of individual, mean, and median values by treatment and study day.

#### 21. GENETIC ANALYSIS

Not applicable.

#### 22. DATA NOT SUMMARIZED OR PRESENTED

The unscheduled visits will not be summarized, but listed.

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final2018-02-07 Document:

Version Number: Final 1.0 Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

Author:




# 23. REFERENCES

Protocol amendment dated 30May2017

Annotated study book Version 2 dated 26Dec2016

APPENDIX 1. **PARTIAL DATE CONVENTIONS** 

Imputed dates will NOT be presented in the listings.

Algorithm for Treatment Emergence of Adverse Events:

| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| | Partial | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| | Missing | If start date < study med start date, then not TEAE |
| | | If start date >= study med start date, then TEAE |
| Partial, but known components show that it cannot be on or after study med start date | Known | Not TEAE |
| | Partial | Not TEAE |
| | Missing | Not TEAE |

\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\\Final2018-02-07 Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005



STATISTICAL ANALYSIS PLAN


| START DATE | STOP DATE | ACTION |
|---|---|---|
| Partial, could be on or after study med start date | Known | If stop date < study med start date, then not TEAE If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e., last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, then not TEAE If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |
| Missing | Known | If stop date < study med start date, then not TEAE If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e., last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, then not TEAE If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |

Algorithm for Prior / Concomitant Medications:

Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Reference: CS\_WI\_BS005

Template No: CS\_TP\_BS016 Revision 4



# STATISTICAL ANALYSIS PLAN


| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known | If stop date < study med start date, assign as prior If stop date >= study med start date assign as concomitant |
| | Partial | Impute stop date as latest possible date (i.e., last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant |
| | Missing | If stop date is missing, it could never be assumed a prior medication, assign as concomitant |
| Partial | Known | Impute start date as earliest possible date (i.e., first day of month if day unknown or 1st January if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant |

Document: Version Number: Final 1.0 Author: Version Date: 07Feb2018

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

24 July 2019



STATISTICAL ANALYSIS PLAN


| START DATE | STOP DATE | ACTION |
|---|---|---|
| | Partial | Impute start date as earliest possible date (i.e., first day of month if day unknown or 1st January if day and month are unknown) and impute stop date as latest possible date (i.e., last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant |
| | Missing | If stop date is missing, it could never be assumed a prior medication, assign as concomitant |
| Missing | Known | If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant |
| | Partial | Impute stop date as latest possible date (i.e., last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant |
| | Missing | Assumed concomitant |

Template No: CS\_TP\_BS016 Revision 4 Reference: CS\_WI\_BS005

Effective Date: 01Apr2016

AnaptysBio Inc. Protocol No: ANB020-003 Version No.1.0



AnaptysBio Inc. PROTOCOL ANB020-003 

24 July 2019

## TABLE SHELLS

Placebo-Controlled Proof of Concept Study to Investigate ANB020 Activity in Adult Patients with Peanut Allergy

Study No. ANB020-003


24 July 2019

| Minuma Com | - |
|------------|-----|
| ⊜IQ\ | /IA |

Table Shells


# Output Templates Signature Page

Table Shells Draft 3.0 (Dated 07Feb2018) for Protocol ANB020-003.

| | Name | Signature | Date | |
|-----------|---------------------|-----------|------|---|
| Author | | | | |
| Position: | | | | |
| Company: | IQVIA <sup>TM</sup> | | | _ |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study

| | Name | Signature | Date |
|---------------------------|---------------------|-----------|-----------|
| Reviewed and Approved By: | | | |
| Position: | | | 11-4-18 |
| Company: | IQVIA <sup>TM</sup> | | |
| Reviewed and Approved By: | | | |
| Position: | | | |
| Company: | ΜΛΙΥ <sub>ΙΜ</sub> | | |
| Reviewed and Approved By: | | | 11 APROOK |
| Position: | | | |

AnaptysBio Inc. Version No.1.0 Protocol No: ANB020-003

24 July 2019




| Company: | IQVIATM |
|---------------------------|----------------------|
| Reviewed and Approved By: | 12 APR 2017 |
| Position: | |
| Сотрану: | IQV LA <sup>TM</sup> |
| Reviewed and Approved By: | 4 |
| Position: | 11 APZ Ze18 |
| Company: | AnaptysBio, Inc. |

24 July 2019

| | | Signature | Date | |
|---|---|---|---|---|
| Anthor | | | | |
| Position: | | | | |
| Соприну: | MALY IN | | 4 | |
| Upon review of this document, t | he undersigned approves this<br>Name | | ethorizing that the content is acceptable for the | reporting of this study. |
| Reviewed and Approved By: | Nunc | Signature | Date | - |
| Administration Approved by: | | | | |
| Position: | | | | |
| Company: | IQVIATK | | | - |
| | - | | | - |
| Reviewed and Approved By: | | | Tr. 4 10 | - |
| Maryamos and Approved By: | | | 11 Apr 2018 | |
| Position: | | | | |
| Сомрану: | XVIA™ | | | 1 |
| | | | | ┪ |
| Reviewed and Approved By: | | | | 7 |
| | | | 11 APR 2018 | |
| Position: | | | | _ |

AnaptysBio Inc. Version No.1.0 Protocol No: ANB020-003 24 July 2019



**Table Shells** 


## List of Reviewers

| Reviewer Name | Position/ Role | Company |
|---------------|----------------|---------------------|
| | | IQVIA <sup>TM</sup> |
| | | IQVIA <sup>TM</sup> |
| | | IQVIA™ |
| | | IQVIA™ |
| | | AnaptysBio, Inc |

Version Number: Final 1.0 Version Date: 07Feb2018



Table Shells


## **Modification History**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| Draft 1 0 | 08 Mar 2017 | | Not Applicable-First Draft |
| Version 1 0 | 16 Mar 2017 | | Addressed client comments |
| Draft 2 0 | 05 Jun 2017 | | Revision based on protocol amendment 2 0 dated 30May2017 |
| Draft 2 0 | 13 Jun 2017 | | Implemented SBR comments |
| Draft 2 0 | 28 Jun 2017 | | Implemented PK comments |
| Draft 2 0 | 25 Jul 2017 | | Implemented MW comments, changes based on protocol amendment 3 0 dated 30Jun2017 |
| Draft 3 0 | 07Feb2018 | | Implemented PK comments |
| Final Copy | 10 Apr 2018 | | Prepared the Final copy for sign off |




**Table Shells** 


## Table of Contents

| Output Templates Signature Page | 2 |
|---|---|
| List of Reviewers | 3 |
| Modification History | 4 |
| Table 14.1.1.1 Patient Disposition – All Patients Screened Set | 6 |
| Table 14.1 2.1 Protocol Deviations – Randomized Analysis Set | 7 |
| Table 14.1.3.1 Demographic Characteristics – Randomized Analysis Set | 8 |
| Table 14.1.3.2 Other Baseline Characteristics – Randomized Analysis Set | 9 |
| Table 14.1.3.3 Baseline Disease Characteristics – Randomized Analysis Set | . 11 |
| Table 14.1 3.4 Serum Pregnancy Test – Randomized Analysis Set | . 13 |
| Table 14.1.4.1 Medical History - Randomized Analysis Set | |
| Table 14.1 5.1 Prior Medications by ATC Level - Safety Analysis Set | . 15 |
| Table 14.1.6.1 Concomitant Medications by ATC Level - Safety Analysis Set | |
| Table 14.1.7.1 Study Medication Exposure – Safety Analysis Set | |
| Table 14.2.1.1 Cumulative Tolerated Peanut Dose (Unit) During BPCFC – Full Analysis Set | . 17 |
| Table 14.2.1.2 Primary Efficacy: Total Cumulative Tolerated Peanut Dose (Unit) During BPCFC at Day 14 - Full | |
| Analysis Set | . 18 |
| Table 14.2.2.1 OFC Symptom Score – Full Analysis Set | |
| Table 14.2.2.2 Secondary Efficacy: OFC Symptom Score at Day 14 – Full Analysis Set | |
| Table 14.2.3.1 Exploratory Efficacy: Total Cumulative Tolerated Peanut Dose (Unit) During BPCFC and OFC Symptons | |
| Score at Day 45 – Full Analysis Set | |
| Table 14.3 1.1 Overview of Adverse Events – Safety Analysis Set | |
| Table 14.3 1.2 TEAE by System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14.3.1.2.1 TEAEs by Preferred Term – Safety Analysis Set | |
| Table 14.3.1.3 Serious TEAEs by System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14.3.1.4 TEAEs Leading to Discontinuation from the Study by System Organ Class and Preferred Term – Safet | |
| Analysis Set | |
| Table 14.3.1.5 TEAEs Leading to Interruption of Study Drug by System Organ Class and Preferred Term – Safety | |
| Analysis Set | . 25 |
| Table 14.3.1.6 TEAEs Leading to Death by System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14.3.1.7 Non TEAEs by System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14.3.1.8 Adverse Events due to BPCFC by System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14 3.2.1 TEAEs by Severity, System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14 3.2.2 TEAEs by Severity, System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14.3.3.1 TEAEs by Relationship to Study Drug, System Organ Class and Preferred Term – Safety Analysis Set | |
| Table 14.3.4.1 Markably Abnormal Laboratory Criteria (Local Lab) – Safety Analysis Set | |
| Table 14 3.4.2 Markably Abnormal Laboratory Criteria (Central Lab) – Safety Analysis SetError! Bookmark | |
| defined. | шос |
| Table 14 3.4.3 Potential Clinically Significant Laboratory Assessments – Safety Analysis Set | 30 |
| Table 14 3.4.4 Laboratory Parameters – Safety Analysis Set. | |
| Table 14.3.4.5 Shifts from Baseline in Clinical Laboratory Results – Safety Analysis Set. | 32 |
| Table 14 3.5.1 12-Lead ECG – Safety Analysis Set. | |
| Table 14.3.5.2 Overall ECG and OT Changes from Baseline – Safety Analysis Set | |
| Table 14.3.6.1 Vital Signs – Safety Analysis Set | |
| Table 14.3.7.1 Spirometry – Safety Analysis Set | |
| Table 14.3.7.2 Ashtma Assessment of Symptom Control – Safety Analysis Set | |
| Table 14.3.8.1 Physical Examination – Safety Analysis Set | |
| Table 14.4.1.1 Summary of Serum Concentration of ANB020 – Pharmacokinetic Analysis Set | |
| Table 14.4.1.1 Summary of Serum Concentration of ANB020 – Pharmacokinetic Analysis Set Table 14.4.1.2 Summary of Pharmacokinetic Parameters of ANB020 – Pharmacokinetic Analysis Set | |
| Table 14.5.1.1 Summary of Pharmacodynamic Endpoints – Pharmacodynamic Analysis Set | |
| Table 14.5.1.1 Summary of Pharmacodynamic Endpoints – Pharmacodynamic Analysis Set | |

24 July 2019



Table Shells


Table 14 1 1 1 Patient Disposition - All Patients Screened Set

| | ANB020 | Placebo | Total |
|---|---|---|---|
| | (N=XX) | (N=XX) | (N=xx) |
| Category | n (%) | n (%) | n (%) |
| Curegory | 11 (70) | 11 (70) | 11(70) |
| Patients in Randomized Analysis Set | xx | xx | xx |
| Patients Administered the Treatment | xx (xx x) | xx (xx x) | xx (xx x) |
| | | | () |
| Patients in FAS Population | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients in SAF Population | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients in PK Analysis Set | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients in PD Analysis Set | xx (xx x) | xx (xx x) | xx (xx x) |
| ,,,,, | () | | ( |
| Patients who Completed the Study | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients who Completed the Study till Day 14 | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients who Completed the Study till Day 45 | xx (xx x) | xx (xx x) | xx (xx x) |
| | () | | |
| Patients who Discontinued the Study | xx (xx x) | xx (xx x) | xx (xx x) |
| Reason for Discontinuation | (, | | |
| Adverse Event | xx (xx x) | xx (xx x) | xx (xx x) |
| Death | xx (xx x) | xx (xx x) | xx (xx x) |
| | AA (AA A) | an (an A) | aa (aa a) |
| Lack of compliance of protocol | xx (xx x) | xx (xx x) | xx (xx x) |
| Other | xx (xx x) | xx (xx x) | xx (xx x) |
| Out. | aa (aa a) | ma (mt n) | ins (ins a) |

Source: Listing 16 1 2 1, 16 1 2 2

- N is the number of patients within each treatment group in the Randomized Analysis Set

- Percentages are based on the number of randomized patients in the respective treatment arm (N)

- Percentage for reason for discontinuation is based on number of patients who discontinued the study

Programming Note (not part of table): Add missing row where necessary Percentage for reason for discontinuation shall be taken from discontinued patients

\\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document: Author:

24 July 2019



Table Shells


Table 14 1 2 1 Protocol Deviations - Randomized Analysis Set

| | | , | |
|---|---|---|---|
| Deviations/Violations | ANB020<br>(N=XX)<br>n (%) | Placebo<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
| Patients with major protocol deviations | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients with category 1 deviation | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients with category 2 deviation | xx (xx x) | xx (xx x) | xx (xx x) |

Source: Listing 16 1 11 1

- N is the number of patients within each treatment group in the Randomized Analysis Set
   Percentages are based on the number of randomized patients in the respective treatment arm (N)
- Patients with multiple protocol deviations within the same category are counted only once under that category

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document: Author:

24 July 2019



Table Shells


Table 14 1 3 1 Demographic Characteristics - Randomized Analysis Set

| Characteristic | Statistics | ANB020<br>(N=XX) | Placebo<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|---|
| Age (years) | n<br>Mean (SD)<br>Median<br>Min, Max | XX<br>XX X (XX XX)<br>XX X<br>XX, XX | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | xx<br>xx x (xx xx)<br>xx x<br>xx, xx |
| Gender<br>Male<br>Female | n (%) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) |
| Child Bearing Potential Females<br>Yes<br>No | n (%) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) |
| If Not Child Bearing Potential,<br><categories></categories> | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Race <categories></categories> | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Ethnicity <categories></categories> | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Weight (Kg) | | | | |
| Height (m) | | | | |
| BMI(kg/m²) | | | | |

Source: Listing 16 1 1 1

Document: \\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

<sup>-</sup> N is the number of patients within each treatment group in the Randomized Analysis Set Percentages are based on the number of randomized patients in the respective treatment arm (N) Programming Note (not part of table): Add missing row where applicable Present descriptive statistics similar to age for weight, height and BMI (present n, mean, SD, min, max, median)

24 July 2019




Table 14 1 3 2 Other Baseline Characteristics - Randomized Analysis Set

| aaracteristic | Statistics | ANB020<br>(N=XX) | Placebo<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|---|
| in Prick Test and ImmunoCAP Testing | | | | |
| Performed Within 8 Weeks of Screening? Yes No | n (%) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) |
| Peanut Extract<br>Done | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Longest Wheal Diameter (mm) | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | XX<br>XX X (XX XX)<br>XX X<br>XX, XX | xx<br>xx x (xx xx)<br>xx x<br>xx, xx |
| Orthogonal Diameter at the Mid-Point of Longest Axis (mm) | | | | |
| Not Done | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Positive Control<br>Done | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Longest Wheal Diameter (mm) | | | | |
| Orthogonal Diameter at the Mid-Point of Longest Axis (mm) | | | | |
| Not Done | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Negative Control<br>Done | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Longest Wheal Diameter (mm) | | | | |
| Orthogonal Diameter at the Mid-Point of Longest Axis (mm) | | | | |

\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document: Author:

24 July 2019



Table Shells


Table 14 1 3 2 Other Baseline Characteristics – Randomized Analysis Set

| | Outer Duscille Citationes | runicolline of runing size see | | |
|---|---|---|---|---|
| Characteristic | Statistics | ANB020 | Placebo | Total |
| | | (N=XX) | (N=XX) | (N=XX) |
| | | (11 222) | (11 222) | (11 222) |
| 37 : P | (0/) | ( ) | | |
| Not Done | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Drugs of Abuse | | | | |
| Sample Collected? | n (%) | | | |
| Yes | 11 (70) | xx (xx x) | xx (xx x) | xx (xx x) |
| Positive | | xx (xx x) | xx (xx x) | xx (xx x) |
| Negative | | xx (xx x) | xx (xx x) | xx (xx x) |
| No | | xx (xx x) | xx (xx x) | xx (xx x) |
| | | () | (-22.14) | () |

Source: Listing 16 1 6 1, 16 1 8 1

### Note:

Document:

Author:

- N is the number of patients within each treatment group in the Randomized Analysis Set
- Percentages are based on the number of randomized patients in the respective treatment arm (N)

Programming Note (not part of table):

- Add missing row where applicable
- Longest Wheal Diameter (mm) and Orthogonal Diameter at the Mid-Point of Longest Axis (mm) will be summariuzed using n, mean, SD, min, max, median

AnaptysBio Inc. Version No.1.0 Protocol No: ANB020-003

24 July 2019



Table Shells


Table 14 1 3 3 Baseline Disease Characteristics – Randomized Analysis Set

| Characteristic | Statistics | ANB020<br>(N=XX) | Placebo<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|---|
| Quantiferon Gold Test [1] | | | | |
| Blood Sample Collected? Yes Positive Negative No | n (%) | xx (xx x)<br>xx (xx x)<br>xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x)<br>xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x)<br>xx (xx x)<br>xx (xx x) |
| Virology | | | | |
| Blood Sample Collected?<br>Yes<br>No | n (%) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) |
| If Yes, Hepatitis B Surface Antigen <categories></categories> | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| Hepatitis C Antibody<br><categories></categories> | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |
| HIV Antibody<br><categories></categories> | n (%) | xx (xx x) | xx (xx x) | xx (xx x) |

Document: \\\ieedc-nas01\a\\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Author:

AnaptysBio Inc. Version No.1.0


24 July 2019



Table Shells


Table 14 1 3 3 Baseline Disease Characteristics - Randomized Analysis Set

| Characteristic | Statistics | ANB020 | Placebo | Total |
|---|---|---|---|---|
| Characteristic | Dietastacs | | 1 Miceoo | |
| | | (NI-VV) | (NI-VV) | (N=XX) |
| | | $(14-\Delta\Delta)$ | $(11-\Delta\Delta)$ | $(1\sqrt{-\Lambda}\Lambda)$ |

Source: Listing 16 1 9 1, 16 1 10 1

Document:

Author:

- N is the number of patients within each treatment group in the Randomized Analysis Set
   Percentages are based on the number of randomized patients in the respective treatment arm (N)
- [1] Test for Tuberculosis

Programming Note (not part of table): Add missing row where applicable This table can be modified as per the data requirement.

\\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Draft\2018-02-07

24 July 2019



Table Shells


Table 14 1 3 4 Serum Pregnancy Test - Randomized Analysis Set

| | Visit | Characteristic | Result | Statistics | ANB020 | Placebo | Total |
|---|---|---|---|---|---|---|---|
| | | | | | (N=XX) | (N=XX) | (N=XX) |
| Serum Pregnancy Test [1] | Baseline | Test Performed | Yes<br>No | n (%) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) |
| | | Outcome | Positive<br>Negative | n (%) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) |
| | < Visits > | | | | | | |

Source: Listing 16 1 5 1

- N is the number of female patients within each treatment group in the Randomized Analysis Set
- Percentages are based on the number of randomized female patients in respective treatment arm (N)
- [1] Only for women of child bearing potential

Programming Note (not part of table): Add missing row where applicable This table can be modified as per the data requirement.

Document: \\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author:

24 July 2019



Table Shells


Table 14 1 4 1 Medical History - Randomized Analysis Set

| System Organ Class<br>Preferred Term | ANB020 | Placebo | Total |
|---|---|---|---|
| rieleited Tellii | (N=XX)<br>n (%) | (N=XX)<br>n (%) | (N=XX)<br>n (%) |
| | 2 (13) | 11(10) | 2 (10) |
| System Organ Class 1 | | | |
| Preferred Term1 | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term2 | xx (xx x) | xx (xx x) | xx (xx x) |
| | xx (xx x) | xx (xx x) | xx (xx x) |
| System Organ Class 2 | | | |
| Preferred Term1 | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term2 | xx (xx x) | xx (xx x) | xx (xx x) |
| | xx (xx x) | xx (xx x) | xx (xx x) |

## Source: Listing 16 1 3 1

Author:

- N is the number of patients within each treatment group in the Randomized Analysis Set
- Patients experiencing multiple events within the same SOC or preferred term are counted only once under those categories
- Percentages are based on the number of randomized patients in the respective treatment arm (N)

Programming Note (not part of table): Number and percentage (%) of patients with Medical History, sorted by decreasing frequency of system organ class and preferred term in total column Mention "Uncoded" if there are any terms which are not coded yet

Document: \\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

24 July 2019



Table Shells


Table 14 1 5 1 Prior Medications by ATC Level - Safety Analysis Set

| | - | | |
|---|---|---|---|
| ATC Level 1 | ANB020 | Placebo | Total |
| ATC Level 3 | (N=XX) | (N=XX) | (N=XX) |
| | n (%) | n (%) | n (%) |
| Number of Patients with at least one Prior Medication | xx (xx x) | xx (xx x) | xx (xx x) |
| ATC Level 1 | xx (xx x) | xx (xx x) | xx (xx x) |
| ATC Level 3 | xx (xx x) | xx (xx x) | xx (xx x) |
| ATC Level 3 | xx (xx x) | xx (xx x) | xx (xx x) |
| *********** | | | |
| | xx (xx x) | xx (xx x) | xx (xx x) |
| ATC Level 1 | xx (xx x) | xx (xx x) | xx (xx x) |
| ATC Level 3 | xx (xx x) | xx (xx x) | xx (xx x) |
| ATC Level 3 | | | |

Source: Listing 16 1 12 1

- N is the number of patients within each treatment group under Safety Analysis Set
- Medications are coded using WHO Drug Dictionary Dec 2016
- Patients with multiple usage of the same medication within the same ATC level 3 term are counted only once
- Percentages are based on number of patients within each treatment group under Safety Analysis Set(N)
- Only the patients with prior medications are summarized

Programming Note (not part of table): Number and percentage (%) of patients with prior medications, sorted by descending order of frequency in total column Add"Uncoded" if any events are not coded yet If ATC level is not present or received from the DM, present this table for only PT's

Programming Note (not part of table): Similar table will be generated as follows:

Table 14 1 6 1 Concomitant Medications by ATC Level - Safety Analysis Set

Tables 14.1.6.1 will be summarized only for patients having atleast one concomitant medication.

Document: \lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author: Version Number: Draft 3.0


24 July 2019



Table Shells


Table 14 1 7 1 Study Medication Exposure – Safety Analysis Set

| | 3100) 1.2001 | cancer and control of the control of | | |
|---|---|---|---|---|
| Charateristic | Statistics | ANB020 | Placebo | Total |
| | | (N=XX) | (N=XX) | (N=XX) |
| | | n (%) | n (%) | n (%) |
| Total Volume Administered | n | xx | xx | xx |
| | Mean (SD) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| | Median | XX X | XX X | XX X |
| | Min, Max | xx, xx | xx, xx | xx, xx |

Source: Listing 16 1 13 1Note:

- N is the number of patients within each treatment group under Safety Analysis Set
- Percentages are based on number of patients within each treatment group under Safety Analysis Set(N)
- IV = Intravenous

Author:

Document: \(\sigma\)\(\text{lieedc-nas01}\(\alpha\)\(\text{biosdata}\)\(\AnaptysBio\)\(\ANB020\)\(\CYA74393\)\(\Biostatistics\)\(\Documentation\)\(\SAP\)\(\Draft\)\(\2018-02-07\)


Version Number: Draft 3.0 Version Date: 07Feb2018



Table Shells

Table 14 2 1 1

| | | Table 14 Z | |
|---|---|---|---|
| | | Cumulative Tolerated Peanut Dose (Unit) I | |
| Visit | Statistics | ANB020 | Placebo |
| | | (N=XX) | (N=XX) |
| Baseline | n | xx | xx |
| Suscinc | Mean (SD) | xx x (xx xx) | xx x (xx xx) |
| | Median | XX X | XX X |
| | Min, Max | XX, XX | XX, XX |
| | IVIIII, IVIAX | AA, AA | AA, AA |
| Day 14 | n | xx | xx |
| | Mean (SD) | xx x (xx xx) | xx x (xx xx) |
| | Median | XX X | XX X |
| | Min, Max | XX, XX | xx, xx |
| Change from Baseline to l | Day 14 n | xx | xx |
| 0 | Mean (SD) | xx x (xx xx) | xx x (xx xx) |
| | Median | XX X | XX X |
| | Min, Max | xx, xx | xx, xx |
| Day 45 | n | xx | xx |
| 24 15 | Mean (SD) | xx x (xx xx) | xx x (xx xx) |
| | Median | XX X | XX X |
| | Min, Max | XX, XX | XX, XX |
| | 171111, 171000 | ഒരു ഒര | aa, aa |
| Change from Baseline to l | Day 45 n | xx | xx |
| | Mean (SD) | xx x (xx xx) | xx x (xx xx) |
| | Median | xx x | xx x |
| | Min, Max | xx, xx | XX, XX |

Source: Listing 16 2 1 1

N is the number of patients within each treatment group under Full Analysis Set
 Baseline is defined as the nearest non-missing value before first dose of study medication

Programming Note: Continue this table for all available visits and respective change from baseline

Document: \\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author:

AnaptysBio Inc. Version No.1.0 Protocol No: ANB020-003

24 July 2019



Table Shells


Table 14 2 1 2
Primary Efficacy: Change from Baseline in Total Cumulative Tolerated Peanut Dose (Unit) During BPCFC at Day 14 – Full Analysis Set

| | Treatment LSMEANS (SE) | Treatment Difference ANB020 vs Placebo | 95% CI for Difference | p-value |
|---|---|---|---|---|
| ANB020 | Placebo | (Standard Error) | | |
| xxxx xxx (xxxx xxx) | XXXX XXX (XXXX XXX) | xxx xx (xxx xxx) | (xxx xx, xxx xx) | 0 xxx |
| Note: | | | | |

- P-value is obtained using ANCOVA model with treatment as fixed effect and baseline value as covariate

Programming Note: Refer SAP for Model

Document: \\\ieedc-nas01\a\\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07\\Author:

Protocol No: ANB020-003 Version No.1.0 24 July 2019



Table Shells


Table 14 2 2 1

| | OFC Sy | mptom Score – Full Analysis Set | |
|---|---|---|---|
| Visit | Statistics | ANB020<br>(N=XX) | Placebo<br>(N=XX) |
| | | (N-AA) | (IV-AA) |
| Baseline (Prior to challenge 1) | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | xx<br>xx x (xx xx)<br>xx x<br>xx, xx |
| Prior to challenge 2 | | | |
| After completion of challenge 1 | | | |
| After completion of challenge 2 | | | |
| 2 hours after the challenge completion | | | |
| Unscheduled time point | | | |
| Day 14 | | | |
| Prior to challenge 1 | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | xx<br>xx x (xx xx)<br>xx x<br>xx, xx |
| Change from Baseline to Prior to<br>challenge 1 of Day 14 | n | xx | xx |
| chanenge 1 of Day 14 | Mean (SD)<br>Median<br>Min, Max | xx x (xx xx)<br>xx x<br>xx, xx | xx x (xx xx)<br>xx x<br>xx, xx |
| Day 45 | | | |
| Day 45<br>Prior to challenge 1 | n<br>Mean (SD)<br>Median | xx<br>xx x (xx xx)<br>xx x | xx<br>xx x (xx xx)<br>xx x |

\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document:

Author:





AnaptysBio Inc. PROTOCOL ANB020-003  Table Shells

Table 14 2 2 1

| | OFC Syn | nptom Score – Full Analysis Set | |
|---|---|---|---|
| Visit | Statistics | ANB020 | Placebo |
| | | (N=XX) | (N=XX) |
| | Min, Max | xx, xx | xx, xx |
| Change from Baseline to time point of Day 45 | n | xx | xx |
| | Mean (SD) | xx x (xx xx) | xx x (xx xx) |
| | Median | xx x | XX X |
| | Min, Max | xx, xx | XX, XX |

Source: Listing 16 2 2 1

- N is the number of patients within each treatment group under Full Analysis Set

- Baseline is defined as the nearest non-missing value before first dose of study medication

Programming Note: Continue this table for all available visits and respective change from baseline

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document: Author:

AnaptysBio Inc. Version No.1.0


24 July 2019




Table Shells

Table 14 2 2 2

| Secondary Emcacy: C | iane from Baseline in OFC Symptom Score at L | Jay 14 – Full Analysis Set | |
|---|---|---|---|
| Treatment LSMEANS (SE) | Treatment Difference ANB020 vs | 95% CI for Difference | p-value |
| Placebo | Placebo | | |
| | (Standard Error) | | |

xxxx xxx (xxxx xxx) xxxx xxx (xxxx xxx) xxx xx (xxx xxx) (xxx xx, xxx xx) 0 xxx

Note:

ANB020

- P-value is obtained using ANCOVA model with treatment as fixed effect and baseline value as covariate

Programming Note: Refer SAP for Model

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document: Author:


61

24 July 2019



Table Shells


Table 14 2 3 1

| | | 20020 21222 | | | |
|---|---|---|---|---|---|
| Change from Baseline in Total Cumulative Tolerated Peanut Dose (Unit) During BPCFC and OFC Symptom Score at Day 45 – Full Analysis Set | | | | | |
| Endpoint | Treatment L | SMEANS (SE) | Treatment Difference ANB020 v | s 95% CI for Difference | p-value |
| | ANB020 | Placebo | Placebo | | |
| | | | (Standard Error) | | |
| Total Cumulative Tolerated Peanut Dose During BPCFC | xxxx xxx (xxxx xxx) | xxxx xxx (xxxx xxx) | xxx xx (xxx xxx) | (xxx xx, xxx xx) | 0 xxx |
| OFC Symptom Score | xxxx xxx (xxxx xxx) | xxxx xxx (xxxx xxx) | xxx xx (xxx xxx) | (xxx xx, xxx xx) | 0 xxx |

### Note:

Document:

Author:

Programming Note: Refer SAP for Model

<sup>-</sup> P-value is obtained using MMRM model with treatment, visit, treatment\*visit as fixed effects and baseline and baseline visit as covariates




Table Shells


Table 14 3 1 1 Overview of Adverse Events - Safety Analysis Set

| Overview of Adverse Events – Safety Analysis Set | | | |
|---|---|---|---|
| Characteristic | ANB020 | Placebo | Total |
| | (N=XX) | (N=XX) | (N=XX) |
| | n (%) | n (%) | n (%) |
| Overall number of TEAEs | XX | XX | XX |
| Overall number of Non-TEAEs | XX | XX | XX |
| Overall number of AE due to BPCFC | XX | XX | XX |
| Number of Patients with at least one | | | |
| TEAE | xx (xx x) | xx (xx x) | xx (xx x) |
| Serious TEAE | xx (xx x) | xx (xx x) | xx (xx x) |
| Severe TEAE | xx (xx x) | xx (xx x) | xx (xx x) |
| Related TEAE | xx (xx x) | xx (xx x) | xx (xx x) |
| Non-TEAE | xx (xx x) | xx (xx x) | xx (xx x) |
| AE due to BPCFC | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients with TEAE by Severity | | | |
| Mild | xx (xx x) | xx (xx x) | xx (xx x) |
| Moderate | xx (xx x) | xx (xx x) | xx (xx x) |
| Severe | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients with TEAE by Final Outcome | | | |
| Recovered | xx (xx x) | xx (xx x) | xx (xx x) |
| Recovering | xx (xx x) | xx (xx x) | xx (xx x) |
| Not Recovered | xx (xx x) | xx (xx x) | xx (xx x) |
| Recovered with Sequelae | xx (xx x) | xx (xx x) | xx (xx x) |
| Fatal | xx (xx x) | xx (xx x) | xx (xx x) |
| Lost to Follow-Up | xx (xx x) | xx (xx x) | xx (xx x) |
| Action Taken with the Study Drug for Patients with TEAE | | | |
| Drug Permanently Discontinued | xx (xx x) | xx (xx x) | xx (xx x) |
| Dose Reduced | xx (xx x) | xx (xx x) | xx (xx x) |
| Dose Interrupted | xx (xx x) | xx (xx x) | xx (xx x) |
| Dose Not Changed | xx (xx x) | xx (xx x) | xx (xx x) |
| None | xx (xx x) | xx (xx x) | xx (xx x) |
| TVOIC | aa (AA A) | AA (AA A) | AA (AA A) |
| Patients with TEAE with Relationship to Study Drug | | | |
| Unrelated | xx (xx x) | xx (xx x) | xx (xx x) |
| Unlikely | xx (xx x) | xx (xx x) | xx (xx x) |

Document:

Author:

24 July 2019




Table Shells

Table 14 3 1 1

| O | verview of Adverse Events – Sa | afety Analysis Set | |
|---|---|---|---|
| Characteristic | ANB020 | Placebo | Total |
| | (N=XX) | (N=XX) | (N=XX) |
| | n (%) | n (%) | n (%) |
| Possible | xx (xx x) | xx (xx x) | xx (xx x) |
| Probable | xx (xx x) | xx (xx x) | xx (xx x) |
| Unknown | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients with TEAE with Seriousness Criteria | | | |
| Death | xx (xx x) | xx (xx x) | xx (xx x) |
| Life-Threatening | xx (xx x) | xx (xx x) | xx (xx x) |
| Inpatient Hospitalization or Prolongation of Existing Hospitalization | xx (xx x) | xx (xx x) | xx (xx x) |
| Persistent or Significant Disability/ Incapacity | xx (xx x) | xx (xx x) | xx (xx x) |
| Congenital Abnormality/ Birth Defect | xx (xx x) | xx (xx x) | xx (xx x) |
| Other Medically Significant Events | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients who Discontinued from the Study Due to TEAE | xx (xx x) | xx (xx x) | xx (xx x) |

Source: Listing 16 3 1 1, 16 3 2 1, 16 3 3 1, 16 3 4 1

Document:

- N is the number of patients within each treatment group under Safety Analysis Set
- Adverse Event terms are coded using latest version of MedDRA
- Patients experiencing multiple events are counted only once within the treatment group
- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)
- AE- Adverse Event, TEAE- Treatment Emergent Adverse Events

Programming Note (not part of table): For count of TEAEs, use the coded term (preferred term)

\\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07





Table Shells


Table 14 3 1 2 TEAE by System Organ Class and Preferred Term - Safety Analysis Set

| ANB020 | ni i | |
|---|---|---|
| | Placebo | Total<br>(N=XX) |
| (N-AA) | (N-AA) | (N-AA) |
| xx (xx x) | xx (xx x) | xx (xx x) |
| xx (xx x) | xx (xx x) | xx (xx x) |
| xx (xx x) | xx (xx x) | xx (xx x) |
| xx (xx x) | xx (xx x) | xx (xx x) |
| xx (xx x) | xx (xx x) | xx (xx x) |
| xx (xx x) | xx (xx x) | xx (xx x) |
| | (N=XX) xx (xx x) xx (xx x) xx (xx x) xx (xx x) xx (xx x) | (N=XX) (N=XX) xx (xx x) xx (xx x) xx (xx x) xx (xx x) xx (xx x) xx (xx x) xx (xx x) xx (xx x) xx (xx x) xx (xx x) |

Source: Listing 16 3 1 1, 16 3 2 1, 16 3 3 1, 16 3 4 1

- N is the number of patients within each treatment group under Safety Analysis Set

- Adverse Event terms are coded using System Organ Class and Preferred term using using latest version of MedDRA
- Patients experiencing multiple events within the same SOC or PT are counted only once under those categories
- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)

## Programming Note (not part of table):

- Table will be sorted in decreasing frequency of system organ class and preferred term of total column Include "Uncoded" if events are not coded A subject can have one or more preferred terms reported under a given system organ class
- Similar tables will be generated for Safety Analysis Set as follows:

Table 14 3 1 2 1 TEAEs by Preferred Term - Safety Analysis Set

Table 14 3 1 3 Serious TEAEs by System Organ Class and Preferred Term - Safety Analysis Set

Table 14 3 1 4 TEAEs Leading to Discontinuation from the Study by System Organ Class and Preferred Term - Safety Analysis Set

Table 14 3 1 5 TEAEs Leading to Interruption of Study Drug by System Organ Class and Preferred Term - Safety Analysis Set

Table 14 3 1 6 TEAEs Leading to Death by System Organ Class and Preferred Term - Safety Analysis Set

Table 14 3 1 7 Non TEAEs by System Organ Class and Preferred Term - Safety Analysis Set

Table 14 3 1 8 Adverse Events due to BPCFC by System Organ Class and Preferred Term - Safety Analysis Set

Document: \lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07






Table Shells


Table 14 3 2 1 TEAEs by Severity, System Organ Class and Preferred Term - Safety Analysis Set

| | | 43 TD 020 | | | 71 1 | |
|---|---|---|---|---|---|---|
| ystem Organ Class | | ANB020<br>(N=XX) | | | Placebo<br>(N=XX) | |
| Preferred Term | Mild | Moderate | Severe | Mild | Moderate | Severe |
| number of Patients with at least one TEAE by Sevenity | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) |
| ystem Organ Class 1 | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term 1 | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term 2 | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) |
| ystem Organ Class 2 | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term 1 | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) | xx (xx x) |

Source: Listing 16 3 1 1, 16 3 2 1, 16 3 3 1, 16 3 4 1

- N is the number of patients within each treatment group under Safety Analysis Set
- Adverse Event terms are coded using System Organ Class and Preferred term using using latest version of MedDRA
- Patients experiencing multiple events within the same SOC or preferred term are counted only once under those categories
- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)
- Patients experiencing the same event with different severity level are counted under the most severe occurrence

## Programming Note (not part of table):

- Table will be sorted in decreasing frequency of system organ class and preferred term of total column Include "Uncoded" if events are not coded
- A subject can have one or more preferred terms reported under a given system organ class

\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document:




Table Shells


Table 14 3 2 1 TEAEs by Severity, System Organ Class and Preferred Term - Safety Analysis Set

| System Organ Class | Total<br>(N=XXX) | | |
|---|---|---|---|
| Preferred Term | Mild | Moderate | Severe |
| Number of Patients with at least one TEAE by Severity | xx (xx x) | xx (xx x) | xx (xx x) |
| System Organ Class 1 | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term 1 | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term 2 | xx (xx x) | xx (xx x) | xx (xx x) |
| System Organ Class 2 | xx (xx x) | xx (xx x) | xx (xx x) |
| Preferred Term 1 | xx (xx x) | xx (xx x) | xx (xx x) |

Source: Listing 16 3 1 1, 16 3 2 1, 16 3 3 1, 16 3 4 1

- N is the number of patients within each treatment group under Safety Analysis Set
- Adverse Event terms are coded using System Organ Class and Preferred term using using latest version of MedDRA
- Patients experiencing multiple events within the same SOC or preferred term are counted only once under those categories
- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)
- Patients experiencing the same event with different severity level are counted under the most severe occurrence

Programming Note (not part of table):

- Table will be sorted in decreasing frequency of system organ class and preferred term of total column Include "Uncoded" if events are not coded
- A subject can have one or more preferred terms reported under a given system organ class

\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document:

Author:

24 July 2019



Table Shells


Table 14 3 3 1
TEAEs by Relationship to Study Drug, System Organ Class and Preferred Term – Safety Analysis Set

| • | | 0, , | , , | |
|---|---|---|---|---|
| | | ANB020 | Placebo | Total |
| System Organ Class | | (N=XX) | (N=XX) | (N=XX) |
| Preferred Term | Related | Not Related | Related Not Related | Related Not Related |
| Number of Patients with at least one TEAE by Relationship | xx (xx x) | xx (xx x) | xx (xx x) xx (xx x) | xx (xx x) xx (xx x) |
| System Organ Class 1 | xx (xx x) | xx (xx x) | xx (xx x) $xx (xx x)$ | xx(xxx) $xx(xxx)$ |
| Preferred Term 1 | xx (xx x) | xx (xx x) | xx (xx x) xx (xx x) | xx(xxx) $xx(xxx)$ |
| Preferred Term 2 | xx (xx x) | xx (xx x) | xx (xx x) xx (xx x) | xx(xxx) $xx(xxx)$ |
| System Organ Class 2 | xx (xx x) | xx (xx x) | xx (xx x) xx (xx x) | xx(xxx) $xx(xxx)$ |
| Preferred Term 1 | xx (xx x) | xx (xx x) | xx (xx x) xx (xx x) | xx (xx x) xx (xx x) |

Source: Listing 16 3 1 1, 16 3 2 1, 16 3 3 1, 16 3 4 1

### Note:

- N is the number of patients within each treatment group under Safety Analysis Set
- Adverse Event terms are coded using System Organ Class and Preferred term using using latest version of MedDRA
- Patients experiencing multiple events within the same SOC or preferred term are counted only once under those categories
- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)
- Patients experiencing the same event with different relationship level are counted under the worst degree of relationship
- AEs with relationship in ("Possible", "Probable" and "Unknown") are mapped to "Related", else to "Unrelated"

## Programming Note (not part of table):

- Table will be sorted in decreasing frequency of system organ class and preferred term of total column Include "Uncoded" if events are not coded
- A subject can have one or more preferred terms reported under a given system organ class

Document: \(\lieedc-nas01\)a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author:

Protocol No: ANB020-003 Version No.1.0 24 July 2019



Table Shells


Table 14 3 4 1 Markably Abnormal Laboratory Criteria (Local Lab) - Safety Analysis Set

| Laboratory Category | Visit | Markably Abnormality | Indication Low/High | ANB020 | Placebo | Total |
|---|---|---|---|---|---|---|
| Parameter | | Criteria | | (N=XX) | (N=XX) | (N=XX) |
| Hematology | | | | | | |
| Parameter 1 | <visits></visits> | Criteria xx | Low | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Criteria xx | Low | xx (xx x) | xx (xx x) | xx (xx x) |
| Parameter 2 | <visits></visits> | Criteria xx | TTI-d. | () | () | () |
| Parameter 2 | Visits | | High | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Criteria xx | High | xx (xx x) | xx (xx x) | xx (xx x) |
| Clinical Chemistry | | | | | | |
| Parameter 1 | <visits></visits> | Criteria xx | Low | xx (xx x) | *** (*** *) | xx (xx x) |
| Parameter 1 | VISIIS | Chiena xx | Low | XX (XX X) | xx (xx x) | xx (xx x) |
| Parameter 2 | <visits></visits> | Criteria xx | High | xx (xx x) | xx (xx x) | xx (xx x) |
| 1 aranku 2 | VISITS | Cincia AA | 1 light | AA (AA A) | AA (AA A) | AA (AA A) |
| Urinalysis | | | | | | |
| Parameter 1 | <visits></visits> | Criteria xx | High | xx (xx x) | xx (xx x) | xx (xx x) |
| | | | | () | () | |
| Parameter 2 | <visits></visits> | Criteria xx | Low | xx (xx x) | xx (xx x) | xx (xx x) |

Source: Listing 16 3 5 1

- N is the number of patients within each treatment group under Safety Analysis Set
   Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)
   Only the incidences of abnormal values according to normal range criteria are summarized

Programming Note (not part of table): Continue this table for

\\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Document: Author:

24 July 2019



Table Shells


Table 14 3 4 2 Potential Clinically Significant Laboratory Assessments - Safety Analysis Set

| Laboratory Category | Visit | Potential Clinical Significance Status | ANB020 | Placebo | Total |
|---|---|---|---|---|---|
| Parameter | | | (N=XX) | (N=XX) | (N=XX) |
| Hematology | | | | | |
| Parameter 1 | <visits></visits> | Normal | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal NCS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal CS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Missing | xx (xx x) | xx (xx x) | xx (xx x) |
| P | 47.40 | N1 | () | () | () |
| Parameter 2 | <visits></visits> | Normal<br>Abnormal NCS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal CS | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) | xx (xx x)<br>xx (xx x) |
| | | Missing | xx (xx x) | xx (xx x) | xx (xx x) |
| Clinical Chemistry | | iviissing | AA (AA A) | an (an a) | aa (aa a) |
| Parameter 1 | <visits></visits> | | | | |
| Urinalysis | | | | | |
| Parameter 1 | <visits></visits> | | | | |

## Urinalysis

Source: Listing 16 3 5 1

- N is the number of patients within each treatment group under Safety Analysis Set

- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)
- NCS Not Clinically Significant, CS Clinically Significant

Programming Note (not part of table): Use all relevant visits and parameters

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document:





Table Shells


Table 14 3 4 3 Laboratory Parameters - Safety Analysis Set

| Visit | Statistics | Actual | ANB020<br>(N=XX)<br>Change from Baseline | | Placebo<br>(N=XX) | | Total<br>(N = XX) |
|---|---|---|---|---|---|---|---|
| Visit | Statistics | Actual | | 1 | (N=XX) | | (N = XX) |
| Visit | Statistics | Actual | Change from Baseline | A 4 1 | | | |
| | | | Change Iron Dascine | Actual | Change from Baseline | Actual | Change from Baselin |
| Baseline | n | XX | - | XX | - | XX | - |
| | Mean (SD) | xx x (xx xx) | - | xx x (xx xx) | - | xx x (xx xx) | - |
| | Median | xx x | - | xx x | - | XX X | - |
| | Min, Max | xx, xx | - | xx, xx | - | XX, XX | - |
| Day 1 | n | xx | xx | xx | xx | xx | xx |
| | Mean (SD) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| | Median | XX X | xx x | XX X | xx x | XX X | XX X |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX | XX, XX |
| Day 45 | | | | | | | |
| ] | Day 1 Day 45 | Mean (SD) Median Min, Max Day 1 n Mean (SD) Median Min, Max Day 45 | Mean (SD) | Mean (SD) | Mean (SD) | Mean (SD) | Median |

Source: Listing 16 3 5 1

- N is the number of patients within each treatment group under Safety Analysis Set
- Baseline is defined as the last non-missing value before first dose of study medication

Programming Note (not part of table): Present all the parameters in Hematology, Clinical Chemistry, and Urinalysis Provide appropriate discreptives for urinalysis Use all relevant visits

\\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Draft\2018-02-07

Document: Author:




24 July 2019




Table 14 3 4 4

| Laboratory Category<br>Parameter | | | Post Baseline Assessments | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline<br>Assessment | ANB020<br>(N=XX) | | | | | | Placebo<br>(N=XX) | | | |
| | Visit | | Low | Normal | High | Missing | Total | Low | Normal | High | Missing | Total |
| Hematology | | | | | | | | | | | | |
| Parameter 1 | Day 1 | Low | XX | xx | XX | xx | XX | XX | xx | XX | xx | XX |
| | | Normal | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | High | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Missing | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Total | xx | XX | xx | XX | xx | XX | xx | XX | XX | XX |
| | Day 2 | | | | | | | | | | | |
| Parameter 2 | | | | | | | | | | | | |

Source: Listing 16 3 5 1

- N is the number of patients within each treatment group under Safety Analysis Set
   Baseline is defined as the last non-missing value before first dose of study medication

Programming Note (not part of table): Present all the parameters in Hematology, Clinical Chemistry and Urinalysis Use all relevant visits

Document: Author:

\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07



24 July 2019




Table Shells

Table 14 3 5 1 12-Lead ECG - Safety Analysis Set

| | | | | ANB020<br>(N=XX) | | Placebo<br>(N=XX) | | Total<br>(N=XX) |
|---|---|---|---|---|---|---|---|---|
| Darameter (Tinit) | Visit | Statistics | Actual | Change from<br>Baseline | Actual | Change from<br>Baseline | Actual | Change from<br>Baseline |
| Parameter (Unit) | VISIT | Stausucs | Actual | Dasenne | Actual | Daseinie | Actual | Daseine |
| Heart Rate (bpm) | Baseline | n | xx | - | xx | - | xx | - |
| | | Mean (SD) | xx x (xx xx) | - | xx x (xx xx) | - | xx x (xx xx) | - |
| | | Median | xx x | - | XX X | - | xx x | - |
| | | Min, Max | xx, xx | - | XX, XX | - | XX, XX | - |
| | Day 45 | n | xx | xx | xx | xx | xx | xx |
| | | Mean (SD) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) | xx x (xx xx) |
| | | Median | XX X | XX X | XX X | XX X | XX X | XX X |
| | | Min, Max | XX, XX | XX, XX | XX, XX | xx, xx | XX, XX | XX, XX |
| PR Interval (msec) | | | | | | | | |
| QRS Interval (msec) | | | | | | | | |
| QT Interval (msec) | | | | | | | | |
| QTc Interval (msec) | | | | | | | | |
| QTcB (msec) | | | | | | | | |
| QTcF (msec) | | | | | | | | |

#### Source: Listing 16 3 6 1

- N is the number of patients within each treatment group under Safety Analysis Set
- Baseline is defined as the nearest non-missing value before first dose of study medication

Programming Note (not part of table): Continue the table for all parameters and all available visits

Document: \\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Author:

Version Number: Draft 3.0 Version Date: 07Feb2018 Version No.1.0







Table Shells


Table 14 3 5 2 Overall ECG and QT Changes from Baseline - Safety Analysis Set

| Category | Visit | Indication | ANB020 | Placebo | Total |
|---|---|---|---|---|---|
| | | | (N=XX) | (N=XX) | (N=XX) |
| Overall Assessment of ECG | Baseline | Nomal | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal NCS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal CS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Missing | xx (xx x) | xx (xx x) | xx (xx x) |
| | | • | | | |
| | Day 45 | Nomal | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal NCS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal CS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Missing | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients reaching a value in QT Interval (msec) at any time | | | | | |
| during treatment above or equal to [1] | ; | >= 450 (msec) | | | |
| duling acadiscin above of equal to | | >= 480 (msec) | | | |
| | | >= 500 (msec) | | | |
| | | 5-500 (HISCC) | | | |
| Patients Experiencing an increase in QT Interval (msec) at | any | >20/ | | | |
| Time During Treatment by more than [1] [2] | | >30 (msec) | | | |
| , | | >60 (msec) | | | |
| Patients Experiencing a decrease in QT Interval (msec) at | any | >30 (msec) | | | |
| Time During Treatment by more than [1] [2] | | , , | | | |
| | | >60 (msec) | | | |

Source: Listing 16 3 6

- N is the number of patients within each treatment group under Safety Analysis Set

- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)
- NCS Not Clinically Significant, CS Clinically Significant
- [1] Cumulative counts, [2] Change from baseline to any observation on treatment

Programming Note (not part of table): Use all relevant visits and parameters

Document: \\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author:


24 July 2019



Table Shells


Table 14 3 6 1 Vital Signs - Safety Analysis Set

| | | | | | NB020<br>N=XX) | | Placebo<br>N=XX) | | Total<br>(N=XX) |
|---|---|---|---|---|---|---|---|---|---|
| Parameter (Unit) | Visit | Time Point | Statistics | Actual | Change from<br>Baseline | Actual | Change from<br>Baseline | Actual | Change from<br>Baseline |
| Pulse Rate (bpm) | <visits></visits> | <time point=""></time> | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | - | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | - | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | - |
| espiratory Rate (resp/min) | <visits></visits> | | | | | | | | |
| ody Temperature (°C) | <visits></visits> | | | | | | | | |
| ody Temperature (°F) | <visits></visits> | | | | | | | | |
| ystolic Blood Pressure (mmHg) | <visits></visits> | | | | | | | | |
| iastolic Blood Pressure (mmHg) | <visits></visits> | | | | | | | | |

#### Source: Listing 16 3 7 1

- N is the number of patients within each treatment group under Safety Analysis Set
- Baseline is defined as the nearest non-missing value before first dose of study medication

Programming Note (not part of table): Continue the table for all parameters and all available visits

Document: \\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author: Version Number: Draft 3.0 Version Date: 07Feb2018 Bio Inc.


24 July 2019



Table Shells


Table 14 3 7 1 Spirometry – Safety Analysis Set

| | | | • | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | | | ANB020<br>(N=XX) | | Placebo<br>(N=XX) | | Total<br>(N=XX) |
| Parameter (Unit) | Visit | Statistics | Actual | Change from<br>Baseline | Actual | Change from<br>Baseline | Actual | Change from<br>Baseline |
| Actual FEV <sub>1</sub> (L) | <visits></visits> | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | - | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | -<br>-<br>- | xx<br>xx x (xx xx)<br>xx x<br>xx, xx | -<br>-<br>- |
| Predicted FEV <sub>1</sub> (L) | <visits></visits> | | | | | | | |
| Percent of Predicted (%) | <visits></visits> | | | | | | | |

Source: Listing 16 3 8 1

Note:

- N is the number of patients within each treatment group under Safety Analysis Set
- Baseline is defined as the nearest non-missing value before first dose of study medication

Programming Note (not part of table): Continue the table for all parameters and all available visits

Document: \(\sigma\)\(\text{lieedc-nas01}\)a\\(\text{biosdata}\)AnaptysBio\\(\text{ANB020}\)\(\text{CYA74393}\)\(\text{Biostatistics}\)\(\text{Documentation}\\(\text{SAP}\)\(\text{Draft}\)\(\text{2018-02-07}\)

Author: Version Number: Draft 3.0


24 July 2019




Table Shells

Table 14 3 7 2 Ashtma Assessment of Symptom Control - Safety Analysis Set

| | | sessing of Symptom Control – Salety Fi | | | |
|---|---|---|---|---|---|
| Category | Visit | Indication | ANB020 | Placebo | Total |
| | | | (N=XX) | (N=XX) | (N=XX) |
| Patients with Asthma Symptoms More than Twice a Week | Baseline | Yes | xx (xx x) | xx (xx x) | xx (xx x) |
| | | No | xx (xx x) | xx (xx x) | xx (xx x) |
| | Day 14 | Yes | xx (xx x) | xx (xx x) | xx (xx x) |
| | Day 14 | No | AA (AA A) | AA (AA A) | AA (AA A) |
| | | 140 | | | |
| Patients Who Woke in Night due to Asthma | <visits></visits> | Yes | xx (xx x) | xx (xx x) | xx (xx x) |
| Patients who woke in Fright due to Astimia | VISIIS | No | xx (xx x) | xx (xx x) | xx (xx x) |
| | | 140 | AA (AA A) | AA (AA A) | AA (AA A) |
| Patients Needed Reliever for Symptoms More than Twice a | | | | | |
| Week | <visits></visits> | | | | |
| wall makes were a care | and the | | | | |
| Patients with Acitivity Limitation due to Asthma | <visits></visits> | | | | |
| Level of Asthma Symptom Control | <visits></visits> | Well Controlled | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Partially Controlled | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Uncontrolled | xx (xx x) | xx (xx x) | xx (xx x) |
| | | | , | | ` ' |

Source: Listing 16 1 7 1

N is the number of patients within each treatment group under Safety Analysis Set
 Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)

Programming Note (not part of table). Use all relevant visits and parameters Table can be modified as per the data requirement

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07 Document:

Author:


24 July 2019



Table Shells


Table 14 3 8 1 Physical Examination – Safety Analysis Set

| Parameter | Visit | Category | ANB020 | Placebo | Total |
|---|---|---|---|---|---|
| | | | (N=XX) | (N=XX) | (N=XX) |
| | | | n (%) | n (%) | n (%) |
| General appearance | Baseline | Normal | xx (xx x) | xx (xx x) | xx (xx x) |
| •• | | Abnormal, NCS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal, CS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Not Done | xx (xx x) | xx (xx x) | xx (xx x) |
| | Day 14 | Normal | xx (xx x) | xx (xx x) | xx (xx x) |
| | , | Abnormal, NCS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Abnormal, CS | xx (xx x) | xx (xx x) | xx (xx x) |
| | | Not Done | xx (xx x) | xx (xx x) | xx (xx x) |
| | Day 45 | | | | |
| | Day 45 | | | | |

Source: Listing 16 3 9 1

Note:

- N is the number of patients within each treatment group under Safety Analysis Set

- Percentages are based on number of patients within each treatment group under Safety Analysis Set (N)

- NCS - Not Clinically Significant, CS - Clinically Significant

Programming Note (not part of table): Continue the table for all other parameters and all available visits May need to add "Missing" row if response is not available for some patients

Document: \(\lieedc-nas01\)a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author: Version Number: Draft 3.0


24 July 2019



Table Shells


Table 14 4 1 1 Summary of Serum Concentration of ANB020 - Pharmacokinetic Analysis Set

| Visit | Nominal Time Point | Statistics | ANB020<br>(N=XX) |
|---|---|---|---|
| Day 1 | Pre-Dose | n, LLOQ(n)<br>Mean (SD)<br>CV<br>Median (Min, Max) | xx, xx<br>xx x (xx xx)<br>xx x<br>xx x (xx, xx) |
| | 0 50 hours post SOI | n, LLOQ (n)<br>Mean (SD)<br>CV<br>Median (Min, Max) | xx, xx<br>xx x (xx xx)<br>xx x<br>xx x (xx, xx) |
| | EOI | | |
| | EOI+3 hours | | |
| Day 2 | 24 hours post SOI | | |
| Day 5 | 96 hours post SOI | | |
| Day 15 | 336 hours post SOI | | |
| Day 45 | 1056 hours post SOI | | |

Source: Listing 16 4 1 1

Document:

- CV = coefficient of variation; EOI = End of Infusion; LLOQ(n) = number of observations ≥ lower limit of quantitation; Max = maximum; Min = minimum; n = number of observations; SD = standard deviation; SOI = Start of Infusion

Programming Note (not part of table): Use all relevant visits and time points

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author:

24 July 2019




Table Shells

Table 14 4 1 2

| | Summary of Pharmacokinetic Parameters of ANB020 – Phan | macokinetic Analysis Set |
|---|---|---|
| Parameter | Statistics | ANB020<br>(N=XX) |
| C <sub>max</sub> | n<br>Mean (SD)<br>CV<br>Median (Min, Max)<br>Gmean (gCV) | xx, xx<br>xx x (xx xx)<br>xx x<br>xx x (xx, xx)<br>xx x (xx xx) |
| t <sub>max</sub> | n<br>Median<br>Min, Max | XX<br>XX XX<br>XX, XX |

Source: Listing 16 4 1 2

Programming Note (not part of table): Continue this for all other summarized parameters, if any

Document: Author:

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2018-02-07

Version Number: Draft 3.0


<sup>-</sup> CV = coefficient of variation; gCV = geometric coefficient of variation; Gmean = geometric mean; Max = maximum; Min = minimum; n = number of observations; SD = standard deviation


24 July 2019



Table Shells


Table 14 5 1 1 Summary of Pharmacodynamic Endpoints - Pharmacodynamic Analysis Set

| | | | | | ANB020<br>(N=XX | | | Placebo<br>(N=XX) | |
|---|---|---|---|---|---|---|---|---|---|
| Analyte (unit) | Visit | Nominal Time Point | Statistics | Observed | Change from<br>Baseline | Relative Change from<br>Baseline (%) | Observed | Change from<br>Baseline | Relative Change from<br>Baseline (%) |
| Serum Cytokines IL-33<br>(unit) | Baseline | - | n | xx | | | xx | | |
| <b>.</b> | | | Mean (SD)<br>Median<br>Min, Max<br>95% CI | xx x (xx xx)<br>xx x<br>xx, xx<br>(xx xx, xx xx) | | | xx x (xx xx)<br>xx x<br>xx, xx<br>(xx xx, xx xx) | | |
| | Day 2 | 24 hours post SOI | n<br>Mean (SD)<br>Median<br>Min, Max<br>95% CI | xx<br>xx x (xx xx)<br>xx x<br>xx, xx<br>(xx xx, xx xx) | xx<br>xx x (xx xx)<br>xx x<br>xx, xx<br>(xx xx, xx xx) | XX<br>XX X (XX XX)<br>XX X<br>XX, XX<br>(XX XX, XX XX) | xx<br>xx x (xx xx)<br>xx x<br>xx, xx<br>(xx xx, xx xx) | xx<br>xx x (xx xx)<br>xx x<br>xx, xx<br>(xx xx, xx xx) | xx<br>xx x (xx xx)<br>xx x<br>xx, xx<br>(xx xx, xx xx) |
| | Day 5 | 96 hours post SOI | | | | | | | |
| | Day 15 | 336 hours post SOI | | | | | | | |
| Leukocytes (unit) | | | | | | | | | |
| Ex Vivo Cytokines <analyte> (unit)</analyte> | | | | | | | | | |

Source: Listing 16 5 1 1, 16 2 5 2, 16 2 5 3

- CI = confidence interval; EOI = End of Infusion; Max = maximum; Min = minimum; n = number of observations; SD = standard deviation; SOI = Start of Infusion

- Relative change from baseline = (actual-baseline)/baseline
- Baseline is defined as the last non-missing value before first dose of study medication

Programming Note (not part of table): Continue the table for all other analytes of Serum Cytokines, Leukocytes, and Ex Vivo peanut antigen challenge cytokines in whole blood at all available visits and respective time points

Document: \\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Draft\2018-02-07

Author:


24 July 2019



Table Shells


Table 14 5 1 2 Statistical Analysis of Pharmacodynamic Endpoints – Pharmacodynamic Analysis Set

| Companison | Parameter | Treatment Difference (Standard Error) | 95% CI | p-value |
|---|---|---|---|---|
| ANB020 vs Placebo | Serum Cytokines IL-33 | xxx xx (xxx xxx) | (xxx xx, xxx xx) | 0 xxx |
| | Serum Cytokines IL-4 | | | |

#### Note:

Programming Note (not part of table): Continue the table for all other analytes of Serum Cytokines, Leukocytes, and Ex Vivo peanut antigen challenge cytokines in whole blood at all available visits and respective time points

Document: \lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draff\2018-02-07 Author:


<sup>-</sup> CI = confidence interval P-value is obtained using Mixed Effect ANCOVA model with treatment, visit, treatment\*visit as fixed effects and baseline value as covariate

AnaptysBio Inc. Protocol No: ANB020-003 Version No.1.0 24 July 2019



Figure Shells


#### FIGURE SHELLS

Placebo-Controlled Proof of Concept Study to Investigate ANB020 Activity in Adult Patients with Peanut Allergy

Study No. ANB020-003

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07

Author: Version Number: Final 1.0

24 July 2019

| - | ar I Car | |
|---|----------|-----|
| = | 101 | /IA |

## Figure Shells

Output Templates Signature Page

Figure Shells Draft 3.0 (Dated 07Feb2018) for Protocol ANB020-003.

| | Name | Signature | Date |
|-----------|---------------------|-----------|-----------|
| Author: | | | DDMMMYYYY |
| Pesition: | | | |
| Company: | JQVIA <sup>TM</sup> | | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---|---|---|---|
| Reviewed and Approved By: | | | DDMMMYYYY |
| Position: | | | |
| Company: | IQVIA <sup>184</sup> | | |
| Reviewed and Approved By: | | | DDMMMYYYY |
| Position: | | | |
| Сотралу: | IQVIATE | | |
| Reviewed and Approved By: | | | DDMMMYYYY<br>11 AYR 20 18 |
| Position: | | | |
| Company: | IQVIA <sup>1M</sup> | | |
| criewed and Approved By: | | | 12 APR 2018 |
| Position: | | | |
| Company: | IQVIA <sup>1N</sup> | | |
| eviewed and Approved By: | | | DDMMMYYYY |
| | | | 1/AFRZ21F |

Document

| Weedc-nas01atbiosdata\AnaptysBlo\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2017-06-28
| Version Number: Final

Version Date:

28JUN20

24 July 2019

| OF H | marr 4 | See | 180 | • | * |
|------|--------|-----|-----|---|---|
| | IC | 1 | 1 | 1 | ٥ |

| Fio | ure | Sh | ells |
|-----|-----|----|------|

#### Output Templates Signature Page

Figure Shells Draft 3.0 (Dated 07Feb2018) for Protocol ANB020-003.

| | Name | Signature | Date |
|-----------|---------------------|-----------|-----------|
| Author: | | | DDMMMYYYY |
| Position: | | | 1 |
| Сотрапу: | IQVIA <sup>IM</sup> | | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study.

| | | DDMMMYYYY |
|---------|---------------------|--------------------------|
| | | 11-4-18 |
| IQVIATM | | |
| | - | DDMMMYYYY |
| IQVIATM | | |
| | | DDMMMYYYY<br>11 APR 2018 |
| IQVIATM | | |
| | | DDMMMYYYY |
| IQVIATM | | |
| | | DDMMMYYYY |
| | IQVIA <sup>TM</sup> | IQVIA <sup>TM</sup> |

Document:

Author:

Final 1.0 Version Number:

Version Date:

28JUN20 17

24 July 2019

| 15.5 | - | howen | - |
|------|----|-------|---|
| 1 | 10 | V | 1 |

# Figure Shells

Output Templates Signature Page Figure Shells Draft 3.0 (Dated 07Feb2018) for Protocol ANB020-003.

| | Name | Signature | Date |
|-----------|---------|-----------|-----------|
| Author: | | | DDMMMYYYY |
| Position: | | | |
| Company: | IQVIAIN | | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is

| | Name | Signature | Date |
|---------------------------|---------------------|-----------|-------------|
| Reviewed and Approved By: | | | DDMMMYYYY |
| Position: | | | |
| Company: | IQVIA <sup>1M</sup> | | |
| Reviewed and Approved By: | | | 11 Apr2018 |
| Position: | | | |
| Company: | IQVIA <sup>1M</sup> | | |
| exiewed and Approved By: | | | DDMMMYYYY |
| Position: | | | 1,, ., . |
| Company: | IÓAIVIM | | |
| viewed and Approved By: | | | DDMMMYYYY |
| Position; | | | |
| Company: | IQVIATM | | |
| ricwod and Approved By; | | | / IAFR ZOIF |

\\leedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2017-06-28 Version Number:

28JUN20 17 Version Date:




AnaptysBio Inc. PROTOCOL ANB020-003  Figure Shells

#### List of Reviewers

| Reviewer Name | Position/ Role | Company |
|---------------|----------------|-----------------|
| | | IQVIA™ |
| | | IQVIA™ |
| | | IQVIA™ |
| | | IQVIA™ |
| | | AnaptysBio, Inc |

Document: \\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07

87

Author: Version Number: Final 1.0 07Feb2018 Version Date:




Figure Shells


#### **Modification History**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| Draft 1 0 | 08 Mar 2017 | | Not Applicable-First Draft |
| Version 1 0 | 16 Mar 2017 | | Addressed client comments |
| Draft 2 0 | 08 Jun 2017 | | Revision based on protocol amendment 2 0 dated 30May2017 |
| Draft 2 0 | 13 Jun 2017 | | Implemented SBR comments |
| Draft 2 0 | 28 Jun 2017 | | Implemented PK comments |
| Draft 2 0 | 25 Jul 2017 | | Implemented MW comments, changes based on protocol amendment 3 0 dated 30Jun2017 |
| Draft 3 0 | 07 Feb 2018 | | Implemented PK comments |

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07




Figure Shells


| Table of Contents | |
|---|---|
| Output Templates Signature Page | . 2 |
| Modification History | . 4 |
| Figure 16.1.7.1 Mean and 95% CI for Between-Treatment Difference in Peanut Dose-Full Analysis Set | . 6 |
| Figure~16.1.7.2~Mean~and~95%~CI~for~OFC~Symptom~Score~by~Treatment~and~Mean~Peanut~Dose~-~Full~Analysis~Set | . 7 |
| Figure 16.1.7.3.1 | . 8 |
| Mean (±SD) Serum Concentration Time Profile of ANB020 After IV infusion – Pharmacokinetic Analysis Set | . 8 |
| Figure 16.1.7.3.2 | . 9 |
| Mean (±SD) Serum Concentration Time Profile of ANB020 After IV infusion – Pharmacokinetic Analysis Set | . 9 |
| $Figure\ 16.1.7.5.1.X\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ infusion-Safety\ Analysis\ Set\dots Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ infusion-Safety\ Analysis\ Set\dots Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ infusion-Safety\ Analysis\ Set\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ infusion-Safety\ Analysis\ Set\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ infusion-Safety\ Analysis\ Set\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ infusion-Safety\ Analysis\ Set\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ infusion-Safety\ Analysis\ Set\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ Individual\ ANB020\ Serum\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profiles\ After\ IV\ Individual\ ANB020\ Serum\ Individual\ ANB020\ Serum\ Individual\ Individual\ ANB020\ Serum\ Individual\ Individ$ | 10 |
| $Figure\ 16.1.7.5.2.X\ Individual\ ANB020\ Serum\ Concentration\ Time\ Profile\ After\ IV\ infusion-Safety\ Analysis\ Set$ | 11 |
| Figure 16.1.7.6 Individual, Median, and Mean Plot of Pharmacodynamic Endpoints - Pharmacodynamic Analysis Set | 12 |

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


Figure Shells


24 July 2019


Figure 16 1 7 1
Mean and 95% CI for Between-Treatment Difference in Peanut Dose–Full Analysis Set



ANB020 - Placebo Peanut dose difference in mg

Source: Table 14 2 1 2, 14 2 3 1

Note: CI = confidence interval Mean difference and 95% CI at Day 14 has been obtained through ANCOVA model with treatment as fixed effect and baseline results as a covariate; and mean difference and 95% CI at Day 45 has been obtained through MMRM ANCOVA model with treatment\*visit as fixed effects and baseline\*visit as covariates

Programmer's Note: Include all possible visits (Baseline, Day 14, Day 45)

Document: \\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2017-07-25 Author:

Version Number: Draft 2.0 Version Date: 25Jul2017



Figure Shells


Figure 16 1 7 2
Mean and 95% CI for OFC Symptom Score by Treatment and Mean Peanut Dose – Full Analysis Set



Source: Table 14 2 2 2, 14 2 3 1

Note: CI = confidence interval Mean at Day 14 has been obtained through ANCOVA model with treatment as fixed effect and baseline results as a covariate; and mean at Day 45 has been obtained through MMRM ANCOVA model with treatment, visit, treatment\*visit as fixed effects and baseline and ba

Programmer's Note: Include all possible visits (Baseline, Day 14, Day 45)
Programmer's Note: Similar plots to be presented for the following parameters

24 July 2019



Figure Shells


Figure~16~1~7~3~1 Mean ( $\pm$ SD) Serum Concentration Time Profile of ANB020 After IV infusion – Pharmacokinetic Analysis Set Linear Scale



Source: Table xxx

Note: SD = standard deviation

End of infusion (EOI) was approximately 1 hour after the start of infusion (SOI)

Document: \\ieedc-nas01a\\biosdata\\AnaptysBio\\ANB020\\CYA74393\\Biostatistics\\Documentation\\SAP\\Draft\\2017-06-28 \\Author:

Version Number: Draft 2.0 Version Date: 28JUN2017

24 July 2019



Figure Shells


Figure~16~1~7~3~2 Mean ( $\pm$ SD) Serum Concentration Time Profile of ANB020 After IV infusion – Pharmacokinetic Analysis Set Semi-logarithmic scale



Source: Table xxx

Document: Author:

Note: SD = standard deviation

End of infusion (EOI) was approximately 1 hour after the start of infusion (SOI)

\\lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Draft\2017-06-28

Version Number: Draft 2.0 Version Date: 28JUN2017






Figure Shells

Figure 16 1 7 5 1 X Individual ANB020 Serum Concentration Time Profiles After IV infusion - Safety Analysis Set Patient 1

Linear Scale



Source: Listing xxx

Programming Note: (not part of table): This plot will be prepared for each subject X will take values from 1-20

\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Draft\2017-06-28 Document: Author:

Version Number: Draft 2.0 Version Date: 28JUN2017





Figure Shells


Figure 16 1 7 5 2 X Individual ANB020 Serum Concentration Time Profile After IV infusion - Safety Analysis Set

Patient 1 Semi-logarithmic scale



Source: Listing xxx

Programming Note: (not part of table): This plot will be prepared for each subject X will take values from 1-20

\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Draft\2017-06-28 Document: Author:

Version Number: Draft 2.0 Version Date: 28JUN2017



Figure Shells


24 July 2019


Figure 16 1 7 6
Individual, Median, and Mean Plot of Pharmacodynamic Endpoints – Pharmacodynamic Analysis Set



Programming Note (not part of table): Present the analytes (by page): Serum Sampling for Biomarkers Serum Cytokines, Leukocytes, Cytokine levels released from pathogenic T cells in the ex vivo whole blood Peanut Challenge Assay Each plot would include a separate postdose presentation (similar to Day 2) for each day an assessment is made per protocol

Document: \\ieedc-nas01a\\biosdata\\AnaptysBio\\ANB020\\CYA74393\\Biostatistics\\Documentation\\SAP\\Draft\\2017-06-28 \\Author:

Version Number: Draft 2.0 Version Date: 28JUN2017


24 July 2019




#### LISTING SHELLS

Placebo-Controlled Proof of Concept Study to Investigate ANB020 Activity in Adult Patients with Peanut Allergy

Study No. ANB020-003


24 July 2019



Listing Shells


## Output Templates Signature Page

Listing Shells Draft 3.0 (Dated 07Feb2018) for Protocol ANB020-003.

| | Name | Signature | Date |
|-----------|---------------------|-----------|-----------|
| Author: | | | DDMMMYYYY |
| Position: | | | |
| Company: | IQVIA <sup>TM</sup> | | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|---------------------------|---------------------|-----------|-----------|
| Reviewed and Approved By: | | | DDMMMYYYY |
| Position: | | | 11-4-18 |
| Company: | IQVIA <sup>TM</sup> | | |
| Reviewed and Approved By: | | | DDMMMYYYY |
| Position: | | | |
| | IQVIATM | | ** |

| Document: | \lieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 |
|---|---|

| AnaptysBio Inc. |
|-----------------|

24 July 2019

Listing Shells


#### Output Templates Signature Page

Listing Shells Draft 3.0 (Dated 07Feb2018) for Protocol ANB020-003.

| | Name | Signature | Date |
|-----------|---------------------|-----------|-----------|
| Author: | | | DDMMMYYYY |
| Position: | | | |
| Company: | IQVIA <sup>TM</sup> | | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study.

| Name | Signature | Date |
|---------|-----------|--------------------------|
| | | DDMMMYYYY |
| IQVIA™ | | |
| | | DDMMMYYYY<br>(1 Apr 2618 |
| | | 1 ((1))1 -0() |
| IQVIATM | 444.4.16 | |
| | IQVIATM | IQVIATM |

| Document | : \\eedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 |
|---|---|

MIOVIA

Listing Shells


| Reviewed and Approved By: | | DDMMMYYYY |
|---------------------------|-------------------|---------------|
| | | 11APR 2018 |
| Position: | | |
| Company: | KJA/Vam | |
| Reviewed and Approved By: | | 12 A? R 2 618 |
| Position: | | |
| Самрыну: | KOVIATH | |
| Reviewed and Approved By: | | DDMMMYYYY |
| | | I I APPLEUR |
| Polition: | | |
| Cumpany: | Anaptyelsio, Inc. | |

Document Weedc-nes01s/bloodsts/AnaptysBloVAHB020xCYA743//3\@iostatistics\Documentation\\$AP\Final(2018-02-07 Author

Version Number: Final 1.0 Version Date: 07Feb2018


24 July 2019




Listing Shells

#### List of Reviewers

| Reviewer Name | Position/ Role | Company |
|---------------|----------------|---------------------|
| | | IQVIA™ |
| | | IQVIA <sup>TM</sup> |
| | | IQVIA <sup>TM</sup> |
| | | IQVIATM |
| | | AnaptysBio, Inc |

\\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 Document:

Author: Version Number: Final 1.0 Version Date: 07Feb2018


24 July 2019




Listing Shells

#### **Modification History**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| Draft 1 0 | 08 Mar 2017 | | Not Applicable-First Draft |
| Version 1 0 | 16 Mar 2017 | | Addressed client comments |
| Draft 2 0 | 05 Jun 2017 | | Revision based on protocol amendment 2 0 dated 30May2017 |
| Draft 2 0 | 13 Jun 2017 | | Implemented SBR comments |
| Draft 2 0 | 28 Jun 2017 | | Implemented PK comments |
| Draft 2 0 | 25 Jul 2017 | | Implemented MW comments, changes based on protocol amendment 3 0 dated 30Jun2017 |
| Draft 3 0 | 07 Feb 2018 | | Implemented PK comments |
| Final 1 0 | 10 Apr 2018 | | Finalized the document for sign off |
| | • | | |

Document: \\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07

Author: \\Version N

Version Number: Final 1.0


24 July 2019



# IMS Health & Quintiles are now

## Listing Shells

| Table of Contents | |
|---|---|
| Output Templates Signature Page | 2 |
| List of Reviewers | 4 |
| Modification History | |
| Listing 16.2.1.1 Patient Screening Summary - All Patients Screened | 8 |
| Listing 16.2.1.2 Patient Disposition - All Patients Screened | 9 |
| Listing 16.2.2 Protocol Deviation - All Patients Screened. | |
| Listing 16.2.3.1 Study Eligibility Criteria - All Patients Screened | |
| Listing 16.2.4.1 Demographic Characteristics - Randomized Analysis Set. | 12 |
| Listing 16.2.4.2 Medical History Diagnosis - Randomized Analysis Set | 13 |
| Listing 16.2.4.3 Serum Pregnancy Test - Randomized Analysis Set | 14 |
| Listing 16.2.4.4 Skin Prick Test and ImmunoCAP Testing - Randomized Analysis Set | 15 |
| Listing 16.2.4.5 Global Initiative for Asthma Assessment of Symptom Control - Randomized Analysis Set | 16 |
| Listing 16.2.4.6 Drug Abuse - Randomized Analysis Set | 17 |
| Listing 16.2.4.7 Virology - Randomized Analysis Set. | 18 |
| Listing 16.2.4.8 TB screening - Randomized Analysis Set | 19 |
| Listing 16.2.4.9 Prior and Concomitant Medications - Safety Analysis Set | |
| Listing 16.2.5.1 Exposure to Investigational Product – Safety Analysis Set | 21 |
| Listing 16.2.6.1 Oral Peanut Food Challenge (BPCFC) - Full Analysis Set | |
| Listing 16.2.6.2 Oral Food Challenge Symptom Scoring - Full Analysis Set. | 23 |
| Listing 16.2.7.1 Treatment Emergent Adverse Events - Safety Analysis Set | |
| Listing 16.2.7.2 Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug - Safety Analysis Set | 25 |
| Listing 16.2.7.3 Serious Treatment Emergent Adverse Events - Safety Analysis Set | |
| Listing 16.2.7.4 Treatment Emergent Adverse Events Leading to Death - Safety Analysis Set | 27 |
| Listing 16.2.7.5 Adverse Events Due to BPCFC - Safety Analysis Set | |
| Listing 16.2.8.1 Clinically Significant Laboratory Results - Safety Analysis Set | |
| Listing 16.2.8.2 ECG - Safety Analysis Set | 30 |
| Listing 16.2.8.3 Vital Signs - Safety Analysis Set | 31 |
| Listing 16.2.8.4 Spirometry - Safety Analysis Set | 32 |
| Listing 16.2.8.5 Physical Examination Results - Safety Analysis Set | |
| Listing 16.2.8.6 Individual ANB020 Serum Concentrations - Safety Analysis Set. | |
| Listing 16.2.8.7.1 Individual ANB020 Serum Pharmacokinetic Parameters - Safety Analysis Set | 35 |
| Document: \\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07 | |
| • | |


24 July 2019




| Lieting Shalle |
|----------------|
| Listing Oriens |

| Listing 16.2.8.7.2 Individual Lambda-z Related Parameters for ANB020 - Safety Analysis Set | 3 |
|---|---|
| Listing 16.2.8.8 Circulating Serum Cytokines - Safety Analysis Set | 3 |
| Listing 16.2.8.9 Leukocytes (Whole Blood) - Safety Analysis Set. | 3 |
| Listing 16.2.8.10 Ex vivo Peanut Challenge Assay for Cytokines Released from T-cells (Whole Blood) - Safety Analysis Set | 30 |
| Listing 16.2.8.11.1 Subjects Excluded from the Pharmacokinetic Analysis Set | 4 |
| Listing 16.2.8.11.2 Data Excluded from the Pharmacokinetic Analysis Set | 4 |

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019

AnaptysBio Inc.

PROTOCOL ANB020-003 



Listing Shells

Listing 16 2 1 1
Patient Screening Summary - All Patients Screened

| Patient No | Treatment | Age/Gender | Date and Time<br>of ICF | Confirmed Informed<br>Consent at Day 1/If<br>No, Specify | Completed study? | If No, Reason for<br>Discontinuation |
|---|---|---|---|---|---|---|
| XXX | XXX | 32/Male | DDMMMYYY<br>YTHH:MM | Yes | Yes | - |
| XXX | XXX | 31/Female | DDMMMYYY<br>YTHH:MM | Yes | No | Screen Failure |
| XXX | XXX | 28/Female | DDMMMYYY<br>YTHH:MM | No: xxxx | No | Subject Withdrew<br>Consent |

Programming Note (not part of table): Sort by patient number, date and time of ICF


24 July 2019




Listing Shells

Listing 16 2 1 2 Patient Disposition - All Patients Screened

| | | | | | Disposition 1221 | | | |
|---|---|---|---|---|---|---|---|---|
| Patient No | Treatment | Age/Gender | Administered the<br>Treatment | Included in<br>Randomized Analysis<br>Set | Included in FAS | Included in SAF | Included in PK<br>Analysis Set | Included in PD<br>Analysis Set |
| XXX | XXX | 32/Male | Yes | Yes | Yes | Yes | Yes | Yes |
| XXX | XXX | 31/Female | | | | | | |
| XXX | XXX | 28/Female | | | | | | |

- 1. All patients who have received at least one dose of ANB020 or placebo and provide at least one evaluable post dose PD measurement without any events or protocol deviation deemed to affect PD assessment.
- 2. All patients who have received ANB020 and have at least one post dose serum concentration data value available for ANB020 without any events or protocol deviation deemed to affect PK assessments.

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019




Listing Shells

Listing 16 2 2
Protocol Deviation - All Patients Screened

| Patient No | Treatment | Age/Gender | Significance | Deviation Date | Deviation Category | Deviation Description | Lead to Patient Exclusion from<br>PK Population | Lead to Patient Exclusion<br>from PD Population |
|---|---|---|---|---|---|---|---|---|
| xxx | XXX | 32/Male | Major | DDMMMYYYY | xxxxxx | xxxxxxxxxxx | Yes | No |
| xxx | xxx | 31/Female | Major | DDMMMYYYY | xxxxxxx | xxxxxxxxxxx | xx | xx |
| xxx | xxx | 28/Female | | | | | | |







Listing 16 2 3 1 Study Eligibility Criteria - All Patients Screened

| Patient No | Age/<br>Gender | Did the patientt meet the eligibility criteria for the study? | If No, Specify criteria |
|---|---|---|---|
| XXX | 32/ | Yes | |
| | Male | | |
| XXX | 31/ | Yes | |
| | Female | | |
| XXX | 28/ | No | INCD7 |
| | Female | | |

Programming Note (not part of table): Sort by patient number

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07 Document:


24 July 2019





Listing Shells

Listing 16 2 4 1
Demographic Characteristics - Randomized Analysis Set

| Patient No /<br>Treatment | Age/Gender | Ethnicity | Race | Weight (Kg) | Height (Kg) | BMI(kg/m²) | If Female, then<br>WOCBP | If Not WOCBP,<br>then Method<br>Used |
|---|---|---|---|---|---|---|---|---|
| XXX/ | 32/Male | xxxxxx | xxxxxx | xx xx | xx xx | xx xx | - | - |
| XXX | | | | | | | | |
| XXX/ | 31/Female | xxxxxx | xxxxxx | xx xx | xx xx | xx xx | Yes | - |
| XXX | | | | | | | | |
| XXX/ | 28/Female | xxxxxx | Xxxxxx | xx xx | xx xx | xx xx | No | Other: xxxx |
| XXX | | | | | | | | |
| Note: | | | | | | | | |
| WOCBP: Women of Chi | ld Bearing Potential | | | | | | | |

Programming Note (not part of table): Sort by patient number; USUBJID may be modified later


24 July 2019

IM5 Health & Quintiles are now


Listing Shells

Listing 16 2 4 2 Medical History Diagnosis - Randomized Analysis Set

| Patient No /<br>Treatment | Age/Gender | Medical History<br>Number | Medical History<br>Diagnosis | Primary System<br>Organ Class | Preferred Term | Start Date/<br>End Date | Currently taking medication? |
|---|---|---|---|---|---|---|---|
| XXX/<br>XXX | 32/Male | xxxx | XXXX | XXXX | xxxx | DDMMMYYYY/<br>DDMMMYYYY | No |
| XXX/<br>XXX | 31/Female | xxxx | XXXX | | | DDMMMYYYY/<br>Ongoing | Yes |
| XXX/<br>XXX | 28/Female | XXXX | XXXX | | | DDMMMYYYY/<br>Ongoing | Yes |

Note: Only patients with relevant medical history have been listed

Programming Note (not part of table): Sort by patient number, medication history number, start date

 $\label{locument:sapking} Document: $$ \underline{\arraycolor: NB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 } $$ $$ \underline{\arraycolor: NB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 } $$ $$ \underline{\arraycolor: NB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 } $$ $$ \underline{\arraycolor: NB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 } $$ $$ \underline{\arraycolor: NB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 } $$ $$ \underline{\arraycolor: NB020\CYA74393\Biostatistics\Documentation\SAP\Final\Arraycolor: NB020\CYA74393\Biostatistics\Documentation\Biostatistics\Biosta$ 


24 July 2019

AnaptysBio Inc.




Listing 16 2 4 3 Serum Pregnancy Test - Randomized Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender | Visit | Was the serum pregnancy test performed? | If No, Specify reason | Date of serum pregnancy test | Result |
|---|---|---|---|---|---|---|
| XXX/ | 32/ | Baseline | Yes | - | DDMMMYYYY | Negative |
| XXX | Female | | | | | |
| | | Day 14 | Yes | - | | |
| | | Day 15 | Yes | - | | |
| XXX/ | 31/ | | No | Xxxx | | |
| XXX | Female | | | | | |
| XXX/ | 28/ | | Yes | | DDMMMYYYY | Positvie |
| XXX | Female | | | | | |

Note: The listings consists only female patients in RND population Programming Note (not part of table): Sort by patient number, date


24 July 2019




Listing 16 2 4 4
Skin Prick Test and ImmunoCAP Testing - Randomized Analysis Set

| Patient<br>No /<br>Treatment | Age/<br>Gender | Was Skin<br>prick test and<br>ImmunoCAP<br>testing<br>performed<br>within 8<br>weeks before<br>screening? | If No,<br>Specify<br>reason | Date and time<br>of test | Peanut<br>extract | Longest<br>wheal<br>diameter<br>(mm) | Orthogonal<br>diameter at<br>the mid-<br>point of the<br>longest axis<br>(mm) | If Not<br>Done,<br>Specify<br>reason | Positive<br>control | Longest<br>wheal<br>diameter<br>(mm) | Orthogonal<br>diameter at the<br>mid-point of<br>the longest<br>axis<br>(mm) | If Not<br>Done,<br>Specify<br>reason | Negative<br>control | Longest<br>wheal<br>diameter<br>(mm) | Orthogonal<br>diameter at the<br>mid-point of<br>the longest<br>axis<br>(mm) | If Not<br>Done,<br>Specify<br>reason |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/<br>XXX | 32/<br>Male | Yes | | DDMMMYYY<br>Y/ hh:mm | Done | xxx | xxx | | Done | xxx | xxx | | Done | xxx | xxx | |
| XXX/<br>XXX | 31/<br>Female | No | xxxx | | Not<br>Done | | | xxx | Not<br>Done | | | xxx | Not Done | | | xxx |
| XXX/<br>XXX | 28/<br>Female | Yes | | DDMMMYYY<br>Y/ hh:mm | Done | xxx | xxx | | Done | xxx | xxx | | Done | xxx | xxx | |

Programming Note (not part of table): Sort by patient number


24 July 2019

AnaptysBio Inc.


IM5 Health & Quintiles are now **AIVOI** Listing Shells

> Listing 16 2 4 5 Global Initiative for Asthma Assessment of Symptom Control - Randomized Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender | Daytime asthma symptoms more than twice a week? | Any night waking due to asthma? | Reliever needed for symptoms more than twice a week? | Any activity limitation due to asthma? | Level of Asthma Symptom<br>Control |
|---|---|---|---|---|---|---|
| XXX/XXX | 32/ | No | No | No | No | Well-controlled (None of these) |
| | Male | | | | | |
| XXX/XXX | 31/ | Yes | Yes | No | No | Partially controlled (1-2 of these) |
| | Female | | | | | |
| XXX/XXX | 28/ | No | No | Yes | Yes | Uncontrolled (3-4 of these) |
| | Female | | | | | |

Programming Note (not part of table): Sort by patient number

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07 Document:


24 July 2019

AnaptysBio Inc.




Listing 16 2 4 6

| Patient No /<br>Treatment | Age/<br>Gender | Visit | Was a sample collected for drugs of abuse? | If No, Specify reason | Date of sample collection | Result | If positive, Specify |
|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male | Baseline | Yes | | DDMMMYYYY | Negative | |
| | | Day 14 | Yes | | DDMMMYYYY | Negative | |
| | | Day 15 | Yes | | DDMMMYYYY | Negative | |
| XXX/XXX | 31/<br>Female | | No | xxxx | | | |
| | 28/<br>Female | | Yes | | DDMMMYYYY | Positvie | xxxx |

Drug Abuse - Randomized Analysis Set

Programming Note (not part of table): Sort by patient number Continue for all other available visits. This listing can be modified as per the data requirement

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07 Document:


24 July 2019




Listing Shells

Listing 16 2 4 7 Virology - Randomized Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender | Was the sample collected? | If No, Specify<br>reason | Date of sample collection | Hepatitis B Surface<br>Antigen | If Not Done,<br>Specify<br>reason | Hepatitis C<br>Antibody | If Not Done ,<br>Specify reason | HIV Antibody | If Not Done ,<br>Specify reason |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male | Yes | | DDMMMYYYY/<br>hh:mm | Negative | | Positvie | | Positvie | |
| XXX/XXX | 31/<br>Female | No | xxxx | | | | | | | |
| XXX/XXX | 28/<br>Female | Yes | | DDMMMYYYY | Positvie | | Negative | | Negative | |

Programming Note (not part of table): Sort by patient number

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07 Document:


24 July 2019

AnaptysBio Inc.




Listing Shells

Listing 16 2 4 8 TB screening - Randomized Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender | Was a blood sample collected for quantiferon gold test? | If No, Specify reason | Date of sample collection | Result |
|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male | Yes | | DDMMMYYYY | Negative |
| XXX/XXX | 31/<br>Female | No | XXXX | | |
| XXX/XXX | 28/<br>Female | Yes | | DDMMMYYYY | Positvie |

Programming Note (not part of table): Sort by patient number

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019

IM5 Health & Quintiles are now **AIVOI** Listing Shells


Listing 16 2 4 9 Prior and Concomitant Medications - Safety Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender | Medication<br>Number | Medication Name<br>Reported/ Preferred Term | Start Date/ End Date/ Ongoing | Dose (Unit)/<br>Frequency/ Route | Indication | Prior or<br>Concomitant |
|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male | 1 | xxxx | DDMMMYYYY/<br>DDMMMYYYY | XXX mg | XXXX | Concomitant |
| XXX/XXX | 31/<br>Female | 2 | xxxx | DDMMMYYYY/<br>DDMMMYYYY | XXX mcg | xxxx | Prior |
| XXX/XXX | 28/<br>Female | 3 | xxxx | DDMMMYYYY/<br>DDMMMYYYY | XXX ml | xxxx | Prior |

Programming Note (not part of table): Sort by patient number, medication number, start date

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\\Documentation\SAP\\Final\2018-02-07 Document:


24 July 2019




#### Listing 16 2 5 1 Exposure to Investigational Product - Safety Analysis Set

| Patient No /<br>Treatment | Age/Gender | IP administered via IV/ If<br>No, reason | Start Date and Start Time | End Date and End Time | Total Volume<br>Administered<br>(mL) | If Total volume<br>administered <100<br>ml, Reason |
|---|---|---|---|---|---|---|
| XXX/XXX | 32/Male | Yes | DDMMMYYYYThh:mm | DDMMMYYYYThh:mm | XXXX | xxxx |
| XXX/XXX | 31/Female | Yes | DDMMMYYYYThh:mm | DDMMMYYYYThh:mm | XXXX | - |
| XXX/XXX | 28/Female | No/ xxxx | | | | |

IP - Investigational Product

IV - Intravenous

Programming Note (not part of table): Sort by patient number, start date, start time

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\\Documentation\SAP\\Final\2018-02-07 Document:


24 July 2019

AnaptysBio Inc.




Listing Shells

Listing 16 2 6 1 Oral Peanut Food Challenge (BPCFC) - Full Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender | Visit | Was oral<br>BPCFC<br>performed? | Cumulative<br>Ingested 1<br>(Unit) | Start Date/<br>Start Time of dose<br>challenge 1 | End Date /<br>End Time of<br>dose<br>challenge 1 | Cumulative<br>Ingested 2<br>(Unit) | Start Date/<br>Start Time of dose<br>challenge 2 | End Date /<br>End Time of<br>dose<br>challenge 2 |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male | Baseline | Yes | XX | DDMMMYYYYTh<br>h:mm | DDMMMYYY<br>YThh:mm | XX | DDMMMYYYYT<br>hh:mm | DDMMMY<br>YYYThh:m<br>m |
| | | Day 14 | | | | | | | |
| | | Day 45 | | | | | | | |
| XXX/XXX | 31/<br>Female | | No | XX | DDMMMYYYYTh<br>h:mm | DDMMMYYY<br>YThh:mm | XX | DDMMMYYYYT<br>hh:mm | DDMMMY<br>YYYThh:m<br>m |
| XXX/XXX | 28/<br>Female | | No | - | - | | | | |

Note: BPCFC=Blind Placebo-Controlled Food Challenge

Programming Note (not part of table): Sort by patient number, start date, start time


24 July 2019




Listing 16 2 6 2

| Patient No /<br>Treatment | Age/<br>Gender | Visit | Time point | Date/ Time of<br>Assessment | Skin Rash/ Pruritus/ Urticaria/<br>Angioedema (Grade) | Nasal Sneezing/ Itching/<br>Congestion/ Rhinorrhea/<br>Airway obstruction (Grade) | Chest Wheezing<br>(Grade) | Abdomen Nausea/<br>Abdominal pain/ Emesis/<br>Diarrhea (Grade) |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male | Baseline Day 14 Day 45 | Prior to<br>challenge 1 | DDMMMYYYY/<br>hh:mm | 3/2/0/3f | 3/2/0/1/3 | 3 | 3/ 2/ 0/ 3<br>3/ 2/ 0/ 3<br>3/ 2/ 0/ 3 |
| XXX/XXX | 31/<br>Female | | Prior to<br>challenge 2 | DDMMMYYYY/<br>hh:mm | 3/2/0/3 | 3/ 2/ 0/ 1/ 3 | 0 | 3/ 2/ 0/ 3 |
| XXX/XXX | 28/<br>Female | | After<br>completion<br>of<br>challenge 2 | DDMMMYYYY/<br>hh:mm | 3/2/0/3 | 3/2/0/1/3 | 3 | 3/2/0/3 |

Programming Note (not part of table): Sort by patient number, start date, start time Continue for all other available visits

Document: \\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019




Listing Shells

Listing 16 2 7 1 Treatment Emergent Adverse Events - Safety Analysis Set

| Patient<br>No /<br>Treatment | Age/<br>Gender/<br>Race | AE<br>Number | System Organ<br>Class/Preferred<br>term/Verbatim<br>Text | Start Date/<br>End Date | Did AE<br>occur prior<br>to the start<br>of IP<br>infusion? | AE<br>Severity | Final<br>Outcome | Action taken<br>with the study<br>drug | Relationship<br>to study drug | Serious/<br>Criteria <sup>[1]</sup> | Did the AE cause<br>the subject to<br>discontinue from<br>the study? | Was subject<br>treated for AE? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | xxxx | xx/xx/xx | DDMMMYYY<br>Y/<br>DDMMMYYY<br>Y | No | Severe | Recovered | Dose interrupted | Unlikely | Yes/ XXX | Yes | No |
| XXX/XXX | 31/<br>Female/<br>Race | xxxx | xx/xx/xx | DDMMMYYY<br>Y/<br>DDMMMYYY<br>Y | Yes | Mild | Fatal | Drug<br>permanently<br>discontinued | Possible | Yes/ XXX | Yes | Yes |
| XXX/XXX | 28/<br>Female/<br>Race | xxxx | xx/xx/xx | DDMMMYYY<br>Y/<br>DDMMMYYY<br>Y | Yes | Moderate | Lost to follow-up | Dose reduced | Probable | No | No | No |

[1] - If SAE led to death, then date of death and primary/ secondary cause of death are provided; if required hospitalization, then date of admission and date of discharge are provided

Programming Note (not part of table): Sort by patient number, AE number, start date

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019




Listing 16 2 7 2 Treatment Emergent Adverse Events Leading to Discontinuation of Study Drug - Safety Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender/<br>Race | AE<br>Number | System Organ<br>Class/Preferred<br>term/Verbatim<br>Text | Start Date/<br>End Date | Did AE occur prior<br>to the start of IP<br>infusion? | AE<br>Severity | Final<br>Outcome | Action taken with<br>the study drug | Relationship<br>to study<br>drug | Serious/<br>Criteria <sup>[1]</sup> | Was subject<br>treated for AE? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | No | Severe | Recovered | Dose interrupted | Unlikely | Yes/ XXX | No |
| XXX/XXX | 31/<br>Female/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Mild | Fatal | Drug permanently<br>discontinued | Possible | Yes/ XXX | Yes |
| XXX/XXX | 28/<br>Female/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Moderate | Lost to<br>follow-up | Dose reduced | Probable | No | Yes |

[1] - If SAE led to death, then date of death and primary/ secondary cause of death are provided; if required hospitalization, then date of admission and date of discharge are provided

Programming Note (not part of table): Sort by patient number, AE number, start date

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019




Listing Shells

Listing 16 2 7 3 Serious Treatment Emergent Adverse Events - Safety Analysis Set

| Patient<br>No /<br>Treatment | Age/<br>Gender/<br>Race | AE<br>Number | System Organ<br>Class/Preferred<br>term/Verbatim<br>Text | Start Date/<br>End Date | Did AE<br>occur prior<br>to the start of<br>IP infusion? | AE<br>Sevenity | Final<br>Outcome | Action taken with<br>the study drug | Relationship<br>to study<br>drug | Seriousness<br>Criteria <sup>[1]</sup> | Did the AE cause<br>the subject to<br>discontinue from<br>the study? | Was subject<br>treated for AE? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | No | Severe | Recovered | Dose interrupted | Unlikely | XXX | Yes | No |
| XXX/XXX | 31/<br>Female/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Mild | Fatal | Drug permanently<br>discontinued | Possible | XXX | Yes | Yes |
| XXX/XXX | 28/<br>Female/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Moderate | Lost to follow-up | Dose reduced | Probable | XXX | No | Yes |

Note:

[1] - If SAE led to death, then date of death and primary/ secondary cause of death are provided; if required hospitalization, then date of admission and date of discharge are provided

Programming Note (not part of table): Sort by patient number, AE number, start date

 $\label{local-prop} \textbf{Document:} $$ \underline{\array} Bio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 $$ $$ \underline{\array} Bio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 $$ $$ \underline{\array} Bio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 $$ $$ \underline{\array} Bio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07 $$ $$ \underline{\array} Bio\ANB020\CYA74393\Biostatistics\B$ 


24 July 2019




Listing 16 2 7 4

Treatment Emergent Adverse Events Leading to Death - Safety Analysis Set

| Gender/<br>Race | Number | System Organ<br>Class/Preferred<br>term/Verbatim Text | Start Date/<br>End Date | Did AE occur prior<br>to the start of IP<br>infusion? | AE<br>Severity | Action taken with<br>the study drug | Relationship<br>to study<br>drug | Cause and<br>Date of Death | Did the AE cause<br>the subject to<br>discontinue from<br>the study? | Was subject<br>treated for AE? |
|---|---|---|---|---|---|---|---|---|---|---|
| 32/<br>Male/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | No | Severe | Dose interrupted | Unlikely | XXX/<br>DDMMMYY<br>YY | Yes | No |
| 31/<br>Female/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Mild | Drug permanently<br>discontinued | Possible | XXX/<br>DDMMMYY<br>YY | Yes | Yes |
| 28/<br>Female/<br>Race | xxxx | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Moderate | Dose reduced | Probable | XXX/<br>DDMMMYY<br>YY | No | Yes |
| 3<br>F<br>F<br>F<br>F | 32/<br>Male/<br>Race<br>31/<br>Female/<br>Race<br>28/<br>Female/ | 32/ XXXX Male/ Race 31/ XXXX Female/ Race 28/ XXXX | 32/ XXXX XX/xx/xx Male/ Race 31/ XXXX XX/xx/xx Female/ Race 28/ XXXX XX/xx/xx Female/ | Male | DDMMMYYYY No | Severe S | DDMMMYYYY No Severe Dose interrupted Male/ Race DDMMMYYYY BII/ XXXX XX/xx/xx DDMMMYYYY Yes Mild Drug permanently discontinued Permale/ Race DDMMMYYYY DDMMMYYYY DDMMMYYYYY DDMMMYYYYY DDMMMYYYYY DDMMMYYYYY DDMMMYYYYY DDMMMYYYYY DDMMMYYYYY DOSE reduced | DDMMMYYYY No Severe Dose interrupted Unlikely | Severe Dose interrupted Unlikely XXX/ XX/xx/xx DDMMMYYYY No Severe Dose interrupted Unlikely XXX/ DDMMMYYY YY YY YY YY Severe Dose interrupted Unlikely XXX/ DDMMMYYYY YY YY YY YY YY | the study? Severe Dose interrupted Unlikely XXX/ Yes |

Programming Note (not part of table): Sort by patient number, AE number, start date


24 July 2019




Listing Shells

# Listing 16 2 7 5 Adverse Events Due to BPCFC - Safety Analysis Set

| Patient<br>No /<br>Treatment | Age/<br>Gender/<br>Race | AE<br>Number | System Organ<br>Class/Preferred<br>term/Verbatim<br>Text | Start Date/<br>End Date | Did AE<br>occur prior<br>to the start of<br>IP infusion? | AE<br>Severity | Final<br>Outcome | Action taken with<br>the study drug | Relationship<br>to study<br>drug | Seriousness<br>Criteria <sup>[1]</sup> | Did the AE cause<br>the subject to<br>discontinue from<br>the study? | Was subject<br>treated for AE? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | No | Severe | Recovered | Dose interrupted | Unlikely | xxx | Yes | No |
| XXX/XXX | 31/<br>Female/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Mild | Fatal | Drug permanently<br>discontinued | Possible | XXX | Yes | Yes |
| XXX/XXX | 28/<br>Female/<br>Race | XXXX | XX/xx/xx | DDMMMYYYY<br>/<br>DDMMMYYYY | Yes | Moderate | Lost to<br>follow-up | Dose reduced | Probable | XXX | No | Yes |

\\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07 Document:


24 July 2019


IM5 Health & Quintiles are now **AIVOI** 

Listing Shells

Listing 16 2 8 1 Clinically Significant Laboratory Results - Safety Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender/<br>Race | Test | Visit | Date | Reference Range | Value[a] | Unit | Change from baseline |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | Hemoglobin | Sreening | DDMMMYYYY | (XX-YY) | xxxx | xx | XXXX |
| XXX/XXX | 31/<br>Female/<br>Race | XXXX | xx | DDMMMYYYY | (XX-YY) | xxxx[H] | xx | xxxx |
| XXX/XXX | 28/<br>Female/<br>Race | xxxx | xx | DDMMMYYYY | (XX-YY) | xxxx[L] | xx | xxxx |

[a] The high (H) or low (L) values are only flagged Programming Note (not part of table): Sort by patient number, test, visit, date Present all the parameters

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\\Documentation\SAP\\Final\2018-02-07 Document:


24 July 2019




Listing Shells

Listing 16 2 8 2 ECG - Safety Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender/<br>Race | 12-Lead ECF<br>Performed? | Date | Visit | Test (Unit) | Value | Change from baseline |
|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | Yes | DDMMMYYYY | Baseline | Heart Rate (bpm) | xxxx | |
| | | | | Day 45 | | xxxx | xxxx |
| | | | | Baseline | PR Interval (msec) | xxxx | xxxx |
| | | | | Day 45 | | | |
| | | | | | QRS Interval (msec) | | |
| | | | | | QTcF (msec) | | |
| XXX/XXX | 31/<br>Female/<br>Race | No/ xxxx | | | | | |

Programming Note (not part of table): Sort by patient number, test, visit, date Present all the parameters for all available visits

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\\Documentation\SAP\\Final\2018-02-07 Document:


24 July 2019



Listing Shells


## Listing 16 2 8 3 Vital Signs - Safety Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender/<br>Race | Vital Signs Collected? | Visit | Test (Unit) | Date and Time | Time Point | Value | Change from baseline |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | Yes | <visits></visits> | Blood Pressure (msec) | DDMMMYYYYTHH:M<br>M | Prior to challenge 1 | xxx/xx | - |
| | | | | | | | Not Done | |
| XXX/XXX | 31/<br>Female/<br>Race | No/ xxxx | | | | | | |

Programming Note (not part of table): Sort by patient number, test, visit, date, time Present all the parameters for all available visits

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019


IMS Health & Quintiles are now

Listing Shells

Listing 16 2 8 4 Spirometry - Safety Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender/<br>Race | Visit | Date | Does subject have<br>a history of<br>asthma? | Predicted FEV1<br>(Unit) | Actual FEV1<br>Measurement<br>(Unit) | Percent of Predicted |
|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | Baseline | DDMMMYYYY | No/ xxxx | | | |
| | | Day 14<br>Day 15 | | | | | |
| | | Day 45 | | | | | |
| XXX/XXX | 31/<br>Female/<br>Race | xx | DDMMMYYYY | Yes | xxxx | xxxx | xxxx |

Programming Note (not part of table): Sort by patient number, test, visit, date

Document: \\ieedc-nas01a\biosdata\AnaptysBio\ANB020\CYA74393\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019




Listing 16 2 8 5 Physical Examination Results - Safety Analysis Set

| Patient No /<br>Treatment | Age/<br>Gender/<br>Race | Visit | Body System | Time point | Date/<br>Time of Assessment | Result | If Abnormal, clinically significant, specify |
|---|---|---|---|---|---|---|---|
| XXX/XXX | 32/<br>Male/<br>Race | Baseline | General appearance | Prior to start of BPCFC | DDMMMYYYYThh:mm | Normal | |
| | | Day 14 | | | | | |
| | | Day 45 | | | | | |
| | | | Head, Eyes, Ears,<br>Nose and Throat | | | | |
| XXX/XXX | 31/<br>Female/ | | | Early termination | DDMMMYYYYThh:mm | Abnormal, clinically significant | xxxx |
| XXX/XXX | Race<br>28/<br>Female/<br>Race | | | Unscheduled time point | DDMMMYYYYThh:mm | Not Done | |

Programming Note (not part of table): Sort by patient number, date, time Present all the Body Systems

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07 Document:


24 July 2019




Listing 16 2 8 6 Individual ANB020 Serum Concentrations - Safety Analysis Set

| Patient No /<br>Treatment | Visit | Nominal Time Point | Blood Sample Collected? If No, Reason | Date and<br>Time | Concentration (Unit) |
|---|---|---|---|---|---|
| XXX/XXX | Day 1 | Pre-Dose | Yes | DDMMMYYYYThh:mm | xxxx |
| | | 0 5 hours post SOI | Yes | DDMMMYYYYThh:mm | xxxx |
| | | EOI | Yes | DDMMMYYYYThh:mm | xxxx |
| | | EOI+3 hours | No: xxxx | - | - |
| XXX/XXX | Day 2 | 24 hours post SOI | | | |
| XXX/XXX | Day 15 | | | DDMMMYYYY/ | xxxx |
| | | | | hh:mm | |

Note:

SOI - Start of Infusion, EOI - End of Infusion

Programming Note (not part of table): Sort by patient number, visit, date, time Present all the visits

Document: \\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019

AnaptysBio Inc.




Listing 16 2 8 7 1 Individual ANB020 Serum Pharmacokinetic Parameters - Safety Analysis Set

| Patient No /<br>Treatment | Cmax (ug/mL) | tmax (h) | AUC(0-last)<br>(h*ug/mL) | AUC(0-inf)<br>(h*ug/mL) | t1/2<br>(h) | Lambda-z<br>(1/h) | CL<br>(L/h) | Vss<br>(L) | Vz<br>(L) |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | xxxx | xxxx | | | | | | | |
| XXX/XXX | xxxx | xxxx | | | | | | | |
| XXX/XXX | xxxx | xxxx | | | | | | | |

Programming Note (not part of table): Sort by patient number, visit All subjects and parameters will be listed

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\\Documentation\SAP\\Final\2018-02-07 Document:


24 July 2019


M5 Health & Quintiles are now

IQVIA

Listing Shells

Listing 16 2 8 7 2 Individual Lambda-z Related Parameters for ANB020 - Safety Analysis Set

| Patient No /<br>Treatment | Lambda-z_lower<br>(h) | Lambda-z_upper<br>(h) | t1/2, Interval<br>(h) | t1/2, N | Rsq | %AUCex<br>(%) |
|---|---|---|---|---|---|---|
| XXX/XXX | | | | | | |
| XXX/XXX | | | | | | |
| XXX/XXX | | | | | | |

Note(s): Lambda-z\_lower = start time (h) of the log-linear regression to determine  $\lambda z$  and t1/2; Lambda-z\_upper = End time (h) of the log-linear regression to determine  $\lambda z$  and t1/2; t1/2, Interval = the time interval in the terminal phase used to determine lambda\_z; t1/2, N = number of observations included in calculation of lambda\_z; ND not determined; Rsq = coefficient of determination for calculation of lambda-z; %AUCex = percentage of AUC(0-inf) extrapolated

Programming Note (not part of table): Sort by patient number, visit All subjects and parameters will be listed

Document: \\ieedc-nas01a\\biosdata\\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019


IMS Health & Quintiles are now **AIVOI** 

Listing Shells

## Listing 16 2 8 8 Circulating Serum Cytokines - Safety Analysis Set

| Patient No /<br>Treatment | Visit | Blood Sample Collected? If No,<br>Reason | Date and<br>Time | Cytokine Analyte (Unit) | Value | Change from<br>Baseline | Relative Change from<br>Baseline |
|---|---|---|---|---|---|---|---|
| XXX/XXX | <visits></visits> | Yes | DDMMMYYYYT/hh:mm | IL-33 (unit) | xxxx | | |
| | <visits></visits> | | | | | | |
| | <visits></visits> | | | | | | |
| | <visits></visits> | | | | | | |

Programming Note (not part of table): Sort by patient number, analyte, visit, date, time Present all the visits where assessment done Present the endpoints Cytokines IL-33, IL-4, IL-5, IL-9, IL-13, sST2

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\\Documentation\SAP\\Final\2018-02-07 Document:


24 July 2019






Listing Shells

## Listing 16 2 8 9 Leukocytes (Whole Blood) - Safety Analysis Set

| Patient No /<br>Treatment | Visit | Blood Sample Collected? If<br>No, Reason | Date and<br>Time of Collection | Date and Time of Sample<br>Run | Value (10E3/uL) | Result | Change from<br>Baseline | Relative Change<br>from Baseline |
|---|---|---|---|---|---|---|---|---|
| XXX/XXX | Baseline | Yes | DDMMMYYYYT<br>hh:mm | DDMMMYYYYT<br>hh:mm | xxxx | Normal | | |
| | Day 2 | Yes | DDMMMYYYYT<br>hh:mm | DDMMMYYYYT<br>hh:mm | xxxx | Abnormal<br>NCS | | |
| | Day 45 | No: xxxx | - | - | | | | |

NCS - Not Clinically Significant, CS - Clinically Significant

Programming Note (not part of table): Sort by patient number, visit, date and time of collection Present all the visits where assessment done

\\lieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\\Documentation\SAP\\Final\2018-02-07 Document:


24 July 2019



Listing Shells


# Listing 16 2 8 10 Ex vivo Peanut Challenge Assay for Cytokines Released from T-cells (Whole Blood) - Safety Analysis Set

| Patient No /<br>Treatment | Visit | Blood Sample Collected?<br>If No, Reason | Date and<br>Time of Collection | Time Stimulated<br>(Hours) | Date and Time of<br>Sample Run | Analyte<br>(Unit) | Value | Change from<br>Baseline | Relative<br>Change from<br>Baseline |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XXX | Baseline | Yes | DDMMMYYYYT<br>hh:mm | Hh:mm | DDMMMYYYYT<br>hh:mm | xxx (unit) | xxxx | | |
| | Day 2 | | | | | | | | |
| | Day 5 | | | | | | | | |
| | Baseline | | | | | xxx (unit) | | | |
| | Day 5 | | | | | | | | |
| | | | | | | xxx (unit) | | | |

Programming Note (not part of table): Sort by patient number, analyte, visit, date and time of collection Present all the visits where assessment done Present all analytes

Document: \\ieedc-nas01a\\biosdata\AnaptysBio\ANB020\CYA74393\\Biostatistics\Documentation\SAP\Final\2018-02-07


24 July 2019




Listing 16 2 8 11 1
Subjects Excluded from the Pharmacokinetic Analysis Set

| Patient No / | |
|---------------------------|-------------------------|
| Patient No /<br>Treatment | Reason(s) for exclusion |


24 July 2019




Listing Shells

# Listing 16 2 8 11 2 Data Excluded from the Pharmacokinetic Analysis Set

| Patient No / | Patient No / | |
|--------------|---------------|-------------------------|
| Treatment | Data excluded | Reason(s) for exclusion |

Document: \(\ieedc-nas01a\)\(\begin{array}{linear} \left\) \(\ieedc-nas01a\)\(\begin{array}{linear} \left\) \(\ieedc-nas01a\)
